# Protocol IRB # Pro00001295

# Tandem Autologous Hematopoietic Stem Cell Transplantation with Melphalan Followed by Melphalan and Bortezomib in Patients with Multiple Myeloma

| Protocol Version: | Date of Protocol |
|-------------------|------------------|
| Original Version | 25Feb2010 |
| Amendment 1 | 03Aug2010 |
| Amendment 2 | 02Nov2010 |
| Amendment 3 | 16Oct2012 |
| Amendment 4 | 29May2013 |
| Amendment 5 | 19Jun2014 |
| Amendment 6 | 17Nov2016 |
| Amendment 7 | 06Jun2018 |
| Amendment 8 | 08Nov2019 |

# BLOOD AND MARROW TRANSPLANTATION PROGRAM HACKENSACK UNIVERSITY MEDICAL CENTER

Principle Investigator:

Michele L. Donato, M.D. (551) 996-5900

# TABLE OF CONTENTS

| 1 | INTR<br>1.1<br>1.2<br>1.3<br>1.4 | ODUCTION AND STUDY RATIONALE Overview of the Disease Melphalan VELCADE (bortezomib) for Injection Combination of Bortezomib and Other Agents | 6<br>6<br>9<br>11<br>15 |
|---|---|---|---|
| 2 | STUI<br>2.1<br>2.2 | OY OBJECTIVES Primary Objective Secondary Objectives | 18<br>18<br>18 |
| 3 | 3.1<br>3.2<br>3.3<br>3.4<br>3.5<br>3.6<br>3.7<br>3.8<br>3.9<br>3.10<br>3.11<br>3.12<br>3.13<br>3.14<br>3.15<br>3.16<br>3.17<br>3.18<br>3.19<br>3.20<br>3.21<br>3.22<br>3.23<br>3.24<br>3.25<br>3.26 | Bortezomib Stem Cell Infusion Post-transplant Cytokine Administration Post-transplant Supportive Care Disease Response. Timing between Transplant Procedures Dosing Agents Pre-Transplant Therapy Treatment Assignment Blinding, Packaging, and Labeling Concomitant Treatment Treatment Compliance Duration of Treatment and Patient Participation | 19 19 19 19 19 19 21 22 23 23 23 23 24 27 27 27 28 28 28 29 29 30 31 31 31 31 32 32 32 |
| 4 | 3.27<br>ADV<br>4.1<br>4.2<br>4.3 | Termination of Treatment and/or Study Participation ERSE EVENTS Definitions Procedures for AE and SAE Reporting Assessment of Toxicity | 32<br>33<br>33<br>34<br>34 |
| 5 | | tical Evaluation Endpoint Secondary endpoints | 36<br>36<br>36 |

| | 5.3 | Accrual, Registration and Follow-up | 36 |
|---|---|---|---|
| | 5.4 | Sample Size and Power Calculations | 37 |
| | 5.5 | Efficacy analysis | 37 |
| | 5.6 | Statistical Hyopthesis | 38 |
| | 5.7 | Primary Endpoint | 38 |
| | 5.8 | Secondary endpoints | 38 |
| | 5.9 | Safety Analysis | 39 |
| | 5.10 | Stopping Rules | 39 |
| | 5.11 | Monitoring Compliance | 40 |
| | 5.12 | Data Management and Analysis | 40 |
| 6 | ADMINISTRATIVE REQUIREMENTS | | |
| | 6.1 | Good Clinical Practice | 41 |
| | 6.2 | Ethical Considerations | 41 |
| | 6.3 | Patient Information and Informed Consent | 41 |
| | 6.4 | Protocol Registration | 41 |
| | 6.5 | Patient Confidentiality | 41 |
| | 6.6 | Record Retention | 42 |
| | 6.7 | Investigation New Drug Exemption | 42 |
| 7 | KAR | NOFSKY PERFORMANCE STATUS SCALE | 43 |
| 8 | BOD | Y SURFACE AREA AND CREATININE CLEARANCE | |
| | CALCULATIONS | | |
| 9 | DECLARATION OF HELSINKI | | |
| 10 | COM | MON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS | 49 |
| 11 | REFE | ERENCES | 49 |

| Abbreviation | Definition |
|--------------|---------------------------------------------------|
| °C | degrees Celsius |
| μM | Micromolar |
| 20S | 20S proteasome subunit |
| AE | adverse event |
| ANC | absolute neutrophil count |
| Bc1-2 | B-cell lymphoma-2; a gene that inhibits apoptosis |
| BSA | body surface area |
| CAM | cell adhesion molecules |

**Abbreviation Definition** 

cm Centimeter

CR Complete Response

CTCAE (NCI) Common Terminology Criteria for Adverse Events

CTEP Cancer Therapy Evaluation Program

dL Deciliter

DLT Dose Limiting Toxicity
DNA deoxyribonucleic acid

FDA Food and Drug Administration

GCP Good Clinical Practice
GLP Good Laboratory Practice

ht Height

IkB I kappa B kinase; cytokine response kinase that activates

transcription factor NF-kappa b at serine 32 and 36

ICAM-1 intercellular adhesion molecule 1

ICH International Conference on Harmonisation

IEC Independent Ethics Committee

IND Investigational New Drug
IRB Institutional Review Board

IV Intravenous

I**\***B ✓ I kappa B alpha-associated protein kinase

kg Kilogram

Ki inhibitory constant

lbs Pounds

m²square metersmgMilligramminMinutemLMilliliter

mm<sup>3</sup> cubic millimeters

mmol Millimole

MTD Maximum Tolerated Dose
NCI National Cancer Institute

NF-KB nuclear factor-KB

| Abbreviation | Definition |
|--------------|----------------------------------------------------------|
| ng | Nanogram |
| nM | Nanomole |
| p21 | p21(ras) farnesyl-protein transferase |
| p27 | cyclin-dependent kinase inhibitor |
| p53 | tumor suppressor protein with molecular weight of 53 kDa |
| SAE | serious adverse event |
| US | United States |
| USP | United States Pharmacopeia |
| VCAM-1 | vascular cell adhesion molecule 1 |
| w/w | weight-to-weight ratio |
| wt | Weight |

#### 1 INTRODUCTION AND STUDY RATIONALE

#### **Background**

#### 1.1 Overview of the Disease

Multiple myeloma is the second most common hematological malignancy, affecting about 55,000 Americans. Limited control of disease can be achieved with conventional dose chemotherapy but randomized studies reported improved response rates for patients who are treated with dose-intense therapy and autologous hematopoietic stem cell (HSC) transplantation. However, most patients who undergo dose-intense therapy will require salvage therapy at a median of two to three years after transplantation. High-dose melphalan (200 mg/m²) appears to be the most effective conditioning regimen but the potentially greater tumor cell kill of dose-intense melphalan in synergistic combination with other drugs is only now being studied.

#### 1.1.1 Multiple Myeloma

Multiple myeloma is a malignancy of plasma cells and belongs in a family of diseases known as plasma cell dyscrasias. It accounts for about 1% of all cancers and 10% of all hematological malignancies. Thus, it is the second most common "blood cancer," affecting approximately 55,000 Americans. The annual incidence is about 20,000 cases; the annual death rate is about 11,000. The median age at diagnosis is 65 years old. The disease is more common in males (1.3 to 1) and the frequency doubles in African-Americans compared to Caucasians.

### 1.1.2 Clinical Studies of High-Dose Therapy of Multiple Myeloma

Standard dose therapy for most plasma cell disorders includes regimens such as low-dose melphalan (32 mg/m²/month) with prednisone. For patients with multiple myeloma, this regimen results in a 40% overall response rate, but few patients achieve a complete remission and the median duration of response is only 2 years. The median survival is in the range of 3 years and few (<15%) survive 5 years. More aggressive chemotherapy regimens, including VAD, VBMCP and M2, induce remissions more quickly but overall survival rates are not substantially improved (Alexanian and Dimopoulos, 1994).

These poor outcomes led many investigators explored high-dose chemotherapy regimens. In 1983, McElwain used melphalan 140 mg/m² without stem cell support as a salvage therapy in nine patients with refractory myeloma and noted all patients responded to treatment with five patients achieving complete biochemical and bone marrow responses (McElwain and Powles, 1983). This observation of dose-response led to a series of phase I/II trials with and without stem cell support in both newly diagnosed and refractory disease (Attal et al., 1992; Harousseau et al, 1995).

A matched-pair analysis by the Arkansas group and SWOG comparing dose-intense with standard-dose therapy demonstrated the benefit of autologous HSC transplantation for the treatment of multiple myeloma (Barlogie et al., 1997). Event-free (49 vs 27 months) and overall survivals (62+ vs 48 months) were improved for patients treated with dose-intense therapy as part of the initial treatment.

A number of randomized studies comparing dose-intense therapy with autologous stem cell support to standard therapy regimens have been conducted. The French Myeloma Intergroup reported a large-scale randomized trial (IFM 90) that randomized two hundred patients to either conventional dose VMCP/VBAP or autologous bone marrow transplantation with melphalan and total body irradiation after four cycles of induction treatment (Attal et al., 1996). The findings were strikingly in favor of the dose-intense approach with improvements in complete response rates (22% vs 5%) and median probabilities of event-free (27 months vs 18 months) and overall-survivals (60+ months vs 37 months). In contrast, the USIG found no difference in overall survival using the same transplant conditioning regimen but a much more intensive "standard" non-transplant chemotherapy regimen (Barlogie et al., 2006). These authors also acknowledged that the combination of melphalan and TBI is now recognized as an inferior transplant regimen. The French group Myelome Autogreffe (MAG) achieved results comparable to the IFM 90 trial; however, there was no significant difference in overall survivals as a result of unexpected prolonged survivals in the chemotherapy arm (Fermand et al., 2005). The Spanish PETHEMA group did not find a statistically significant difference in EFS and OS between chemotherapy and dose-intensive therapy (Blade et al., 2005). However, only

patients who responded (CR: 15%; PR: 68%; MR: 17%) to conventional dose chemotherapy were randomized and patients in the chemotherapy arm were allowed to cross over into the dose-intensive therapy group. The Italian MMSG compared melphalan-prednisone to two courses of melphalan at 100 mg/m<sup>2</sup> with autologous stem cell support (Palumbo et al., 2004). They found significant improvement in CR and EFS in the transplant arm. The Medical Research Council Myeloma VII trial of 407 patients reported similar results for a comparison of six cycles of BCNU, doxorubicin, cyclophosphamide and melphalan to at least three cycles of doxorubicin, vincristine, methylprednisolone, and cyclophosphamide followed by melphalan at 200mg/m<sup>2</sup> and autologous stem cell transplant (Child et al., 2003). This trial deserves special consideration in that it is the most recent of the randomized trials and was carried out in the era of more advanced supportive care and the availability of newer therapeutic agents. It still showed a statistically significant advantage for HDT in terms of CR, EFS and OS. In addition, it did not show any increase in treatment-related mortality relative to conventional therapy. These randomized trials, all of which showed a trend to, or significantly improved results for patients treated with dose-intense therapy, with the support of numerous phase II trials, clearly indicate that dose–intense therapy with autologous HSCT should be offered to appropriate patients as part of their initial treatment. The median EFS is remarkably constant (25-31 months). It is more difficult to analyze OS results since OS partly depends on subsequent salvage therapy. However, median OS was significantly longer in the three studies where differences in EFS were more marked. In all studies, procedure-related death rate was <5% and not greater than that observed with conventional chemotherapy.

Table 1: Randomized Trials Comparing Conventional Chemotherapy vs. High-dose Therapy

| | | | | CR rate (%) | | | Median EFS (m) | | | Median OS (n | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <u>N</u> | <u>Age</u> | MedianF/U | <u>CC</u> | <u>HDT</u> | <u>P</u> | <u>CC</u> | <u>HDT</u> | <u>P</u> | <u>CC</u> | <u>HDT</u> | |
| IFM 90 | 200 | <u>&lt;65</u> | <u>7 yr</u> | <u>5</u> | 22 | <0.001 | <u>18</u> | <u>28</u> | <u>0.01</u> | <u>44</u> | <u>57</u> | 0 |
| MAG91 | | <u>55-6</u> | | | | | | | | | | |
| | <u>190</u> | <u>5</u> | <u>56 m</u> | ΝE | NE | | <u> 19</u> | <u>25</u> | <u>0.05</u> | <u>45</u> | <u>42</u> | 1 |
| <u>PETHEMA</u> | <u>164</u> | <u>≤65</u> | <u>42 m</u> | <u>11</u> | <u>30</u> | 0.002 | <u>34</u> | <u>42</u> | <u>NS</u> | <u>67</u> | <u>65</u> | 1 |
| Italian MMSG | | <u>50-7</u> | | | | | | | | | | |
| | <u> 195</u> | <u>0</u> | <u>2 yr</u> | <u>7</u> | <u> 26</u> | <0.001 | <u>16</u> | <u>28</u> | 0.0036 | <u>43</u> | <u>58+</u> | 0.0 |
| <u>USIG</u> | <u>50</u> | | | <u>15</u> | <u>17</u> | <u>NS</u> | <u>21</u> | <u>25</u> | <u>0.05</u> | <u>53</u> | <u>58</u> | 1 |
| MRC7 | <u>407</u> | <u>&lt;65</u> | <u>42 m</u> | 8 | <u>44</u> | <0.001 | <u> 19.6</u> | <u>31.6</u> | <0.0001 | <u>42</u> | <u>54</u> | <0 |

<u>Abbreviations: CC=conventional chemotherapy, CR=complete remission, EFS=event free survival, HDT=high-dose</u> therapy, OS=overall survival, NE=not evaluated, NS=difference not statistically significant.

# 1.1.3 Tandem Autologous Transplantation as Initial Therapy

About 10 years ago, the Arkansas transplant program showed the feasibility of 2 consecutive autologous transplants (Vesole et al., 1994). They described 42 patients who received two consecutive autologous PBSC transplants using melphalan 200mg/m<sup>2</sup>. In patients that were capable of receiving 2 transplants, the CR rate increased from 24% after the first transplant to 43% after 2 transplants. This experience has now been extended in over 1000 patients with overall complete remission rates of 40% and projected 5 year event-free and overall survivals of 25% and 40% respectively (Desikan et al., 2002). The French Intergroup randomized 399 newly diagnosed myeloma patients under age 60 to single versus tandem transplants (Attal et al., 2003). They found similar CR rates between the two groups (42% single transplant vs. 50% tandem transplant), but superior seven year event-free (10% vs. 20%, P=0.03) and overall survivals (21% vs. 42%, P=0.01) for the tandem transplant group. For patients who did not achieve a very good partial response (less than 90% reduction in serum or urine paraprotein) after one transplant, the improvement in seven year overall survival was more dramatic (11% vs. 43%, P<0.01). These results support tandem autologous transplants for patients with a diagnosis of multiple myeloma who do not show disease progression after the first transplant.

# 1.1.4 Impact of Impaired Renal Function on Dose-Intense Therapies

Many patients with plasma cell dyscrasias have renal impairment as a result of their disease; early studies of dose-intense therapy tended to exclude these patients. However, the favorable characteristics of melphalan permits transplant therapy to be extended to patients with renal impairment including patients with end-stage renal failure (ESFR). Pharmacokinetic studies of melphalan show comparable clearance rates regardless of renal function (Tricot et al., 1996). The Arkansas group compared 42 patients with renal failure (including 19 requiring dialysis) with 84 patients matched for other prognostic features. Regimen-related mortality was 7% for the group with renal impairment compared to 6% for those with normal renal function. Engraftment kinetics and probabilities of event-free and overall survivals were also similar. This group reported a subsequent series involving 81 patients with renal insufficiency that showed no difference in quality of stem cell collection and engraftment, even for patients on dialysis (Badros et al., 2001).

# 1.1.5 Age as a Limiting Factor

The plasma cell disorders strike older populations of patients; multiple myeloma is rare for patients under the age of 40 years. The Arkansas group reported a slight increase in 60-day mortality for patients over the age 65 undergoing transplantation for the treatment of myeloma (8% vs 2%). However, median event-free (1.5 vs. 2.8 years) and overall survivals (3.3 vs. 4.8 years) were statistically similar (Siegel et al., 1999).

Age has also not been found to be a significant predictor of transplant related mortality in other series. An analysis of 383 consecutive transplants at Temple University actually noted poorer survival of younger patients compared to older patients, presumably a result of the willingness of physicians to offer aggressive treatment to younger patients with higher risk disease or co-morbid illnesses (Goldberg et al., 1998). Conflicting data on this subject in at least 14 studies (6 no effect, 8 adverse) point to the need for patient selection criteria other than chronological age.

#### 1.2 Melphalan

# 1.2.1 Melphalan Non-clinical Pharmacology

Melphalan is a bifunctional alkylating agent that acts principally through covalent reactions with DNA, resulting in the formation of drug-DNA adducts with cross-linking of DNA strands (Samuels and Bitran, 1995). Melphalan's cytotoxic effects are related to its concentration and the duration of exposure to melphalan of the cell (Hall and Tilby, 1992). Enhanced repair of DNA interstrand crosslinks may be a mechanism of resistance that develops after prior exposure to this drug (Spanswick et al., 2002). Melphalan is actively transported into cells by the high-affinity L-amino acid transport system; glutamine and leucine compete for carrier uptake and high levels of these amino acids can reduce drug uptake. Other drugs such as tamoxifen, chlorpromazine, and indomethacin can also impair melphalan uptake and accumulation.

#### 1.2.2 Clinical Pharmacokinetics and Pharmacodynamics

Studies of the pharmacokinetics of oral melphalan were complicated by the highly variable absorption of the drug. Moreover, studies of intravenous melphalan have also showed considerable inter-patient variability in plasma clearance. Pinguet et al studied the pharmacokinetics of melphalan administered at a dose of 140 mg/m<sup>2</sup> in combination with other chemotherapeutic agents to 20 patients undergoing autologous PBSC transplantation (Pinguet et al., 1997). The medians time to neutrophil and platelet recoveries were 16 and 14.6 days, and the majority of patients (80%) developed WHO grade 3/4 stomatitis. Plasma concentration profiles were biphasic and fitted with a two-compartment model. The maximal concentration at the end of infusion averaged 7.94±3.73 mg/l (range, 1.65-14.5). The mean elimination half-life and the mean residence time were 83.1±27.1 minutes (range, 51.6-16681) and 98.7±26.9 minutes (range 59.5-166.9), respectively. The volume of distribution averaged 1.00±0.62 l/kg (range 0.46-3.12) and total plasma clearance 548.3±300.0 ml/min/m<sup>2</sup> (range, 218.6-1378.8). Plasma levels were below the limits of detection for all patients by 24 hours after melphalan administration. These authors noted large inter-individual variability of these pharmacokinetic parameters. Total clearance of melphalan was significantly correlated with creatinine clearance (r=0.49, p<0.05). A

relationship between melphalan clearance and renal function was also described by Kergueris et al., but this relationship did not explain the large variation in inter-individual overall clearance of the drug (Kergueris et al., 1994). Similar pharmacokinetic results were reported for 20 pediatric and 10 adult patients treated with melphalan 140 mg/m² as a single agent (infused rapidly over 5 minutes; Gouyette et al., 1986). For the adult patients, the elimination half-life ( $t^{1/2}\beta$ ) was 50±7 minutes for patients treated with 140 mg/m² dose and 41±12 minutes for the higher dose of 180 mg/m². Plasma clearance averaged 525 ml/min/m² at 140 mg/m² and 532 ml/min/m² at 180 mg/m².

Melphalan undergoes hydrolysis in the circulation and the amount cleared by the kidneys is not well defined. However, the toxicity of melphalan (hematological or gastrointestinal) is reported higher for patients with diminished renal function. A study of nine patients given a melphalan dose of 5 mg/m² (four of whom subsequently treated with 220 mg/m²) showed highly variable renal clearance of melphalan with the percentage of dose excreted unchanged in the urine ranging from 2.5% to 92.8% (Reece et al., 1988). These authors speculated that the variation in renal clearance observed for these patients could account for the large variation in plasma clearance observed in all studies of melphalan pharmacokinetics.

### 1.2.3 Clinical Toxicities of Melphalan

Dose-related leukopenia, thrombocytopenia, anemia, usually with nadir 2-3 weeks and with recovery 4-5 weeks after dosing (without HSC support) will occur with moderate melphalan dose schedules. Hematological toxicity is the most prominent serious toxicity associated with the use of high-dose melphalan regimens, with neutrophil counts falling to <100/uL about 7 days after administration. However, initial hematological recovery occurs about 3 to 5 days later for patients given hematopoietic stem cell and cytokine support. About 50% of patients will require blood component (red blood cells and/or platelet) support or will develop neutropenic fevers during the period of marrow hypoplasia.

Dose-related nausea and vomiting beginning 2-4 hrs after dosing, peaking at 12 hrs, and persisting for several days, and delayed nausea and vomiting starting 24-48 hrs after administration and persist for multiple days to 3 or 4 weeks occurs with high doses of melphalan. Stomatitis will occur in most patients can be almost completely prevented by prophylactic cooling of the mouth with ice during the infusion of melphalan. A small proportion of patients will develop diarrhea.

Melphalan is associated with a number of rare complications including: hemolytic anemia, abnormal liver function tests with jaundice, renal insufficiency, atrial fibrillation, pulmonary fibrosis and interstitial pneumonitis, skin hypersensitivity, seizures (described in patients with renal failure receiving melphalan, hyponatremia and SIADH, secondary

leukemia and myelodysplastic syndromes, anaphylaxis (rare), and potentially irreversible sterility.

#### 1.3 **VELCADE** (bortezomib) for Injection

#### 1.3.1 Scientific Background

VELCADE™ (bortezomib) for Injection is a small molecule proteasome inhibitor developed by Millennium Pharmaceuticals, Inc., (Millennium) as a novel agent to treat human malignancies. Bortezomib is currently approved by the United States Food and Drug Administration (US FDA) and it is registered in Europe for the treatment of multiple myeloma patients who have received at least one prior therapy.

By inhibiting a single molecular target, the proteasome, bortezomib affects multiple signaling pathways. The anti-neoplastic effect of bortezomib likely involves several distinct mechanisms, including inhibition of cell growth and survival pathways, induction of apoptosis, and inhibition of expression of genes that control cellular adhesion, migration and angiogenesis. Thus, the mechanisms by which bortezomib elicits its antitumor activity may vary among tumor types, and the extent to which each affected pathway is critical to the inhibition of tumor growth could also differ. Bortezomib has a novel pattern of cytotoxicity in National Cancer Institute (NCI) in vitro and in vivo assays (Adams et al., 1999). In addition, bortezomib has cytotoxic activity in a variety of xenograft tumor models, both as a single agent and in combination with chemotherapy and radiation (Steiner et al., 2001; Teicher et al., 1999; Cusack et al., 2001; LeBlanc et al., 2002; Pink et al., 2002). Notably, bortezomib induces apoptosis in cells that over express bcl-2, a genetic trait that confers unregulated growth and resistance to conventional chemotherapeutics (McConkey et al., 1999).

Bortezomib is thought to be efficacious in multiple myeloma via its inhibition of nuclear factor  $\kappa B$  (NF- $\kappa B$ ) activation, its attenuation of interleukin-6 (IL-6)-mediated cell growth, a direct apoptotic effect, and possibly anti-angiogenic and other effects (Hideshima et al., 2001).

# 1.3.2 Non-clinical Pharmacology

Pharmacokinetic (PK) and pharmacodynamic studies were conducted in the rat and cynomolgus monkey. Upon intravenous (IV) bolus administration, bortezomib displays a rapid distribution phase ( $t\frac{1}{2}\alpha$  <10 minutes) followed by a longer elimination phase ( $t\frac{1}{2}\beta$  5–15 hours). Bortezomib has a large volume of distribution (range 5–50 L/kg). The plasma PK profile is well described by a 2-compartment model.

The pharmacodynamic action of bortezomib is well established and can be measured through an ex vivo assay (20S proteasome activity) (Lightcap et al., 2000). This assay was used to determine the duration of drug effect in lieu of the PK data in the early preclinical toxicology studies as well as to set a guide for dose escalation in humans. Following dosing with bortezomib in the rat and cynomolgus monkey, proteasome inhibition in peripheral blood had a half-life less than 24 hours, with proteasome activity returning to pretreatment baseline within 24 hours in monkey and within 48 to 72 hours in rat after a single dose of bortezomib. Further, intermittent but high inhibition (>70%) of proteasome activity was better tolerated than sustained inhibition. Thus, a twice-weekly clinical dosing regimen was chosen in order to allow return of proteasome activity towards baseline between dose administrations

# 1.3.3 Non-clinical Toxicity

Single-dose IV toxicity studies were conducted with bortezomib in the mouse, rat, dog, and monkey to establish the single-dose maximum tolerated dose (MTD). The MTDs were 0.25 mg/kg (1.5 mg/m<sup>2</sup>) and 0.067 mg/kg (0.8 mg/m<sup>2</sup>) in the 2 most sensitive species, rat and monkey, respectively.

Repeat-dose multi-cycle toxicity studies of 3 and 6 months in the rat and 9 months in the monkey, each with 8-week recovery periods, were conducted to characterize the chronic toxicity of bortezomib when administered by the clinical route and regimen of administration. The MTD in the 6-month rat study was 0.10 mg/kg (0.6 mg/m²) and the key target organs were the gastrointestinal (GI) tract, hematopoietic and lymphoid systems. The MTD in the 9-month monkey study was 0.05 mg/kg (0.6 mg/m²) and the key target organs were the GI tract, hematopoietic and lymphoid systems, peripheral nervous system, and kidney. Full or partial reversibility was observed for each of the toxicities described to date.

In general, the nature of the toxicity of bortezomib is similar across species, and target organs of toxicity in animals have been largely predictive of human toxicity. The toxicity of bortezomib in animals is characterized by a steep dose-response with mortality seen at dosages above the MTD. The cause of death at acutely lethal dosages is considered to be related to indirect cardiovascular (CV) effects of hypotension and vascular changes with secondary bradycardia and the cause of death in long-term studies has been attributed to GI or hematologic toxicity. The pharmacologic effects of bortezomib on the CV system have been extensively characterized and have demonstrated that indirect effects on CV function occur only at acutely lethal dosages and are abrogated by routine supportive care.

Additional detailed information regarding the nonclinical pharmacology and toxicology of bortezomib may be found in the 2006 Investigator's Brochure.

# 1.3.4 Clinical Pharmacokinetics and Pharmacodynamics

The clinical pharmacology characterization of bortezomib has been determined from phase 1 studies in subjects with solid tumors and hematological malignancies, and confirmed in phase 2 studies in subjects with multiple myeloma.

Bortezomib demonstrates multi-compartmental pharmacokinetics. Following intravenous administration of 1.0 mg/m² and 1.3 mg/m² dose, the mean first-dose maximum observed plasma concentrations of bortezomib were 57 and 112 ng/mL, respectively in 11 patients with multiple myeloma and creatinine clearance values >50 mL/min participating in a pharmacokinetics study. In subsequent doses, mean maximum observed plasma concentrations ranged from 67 to 106 ng/mL for the 1.0 mg/m² dose and 89 to 120 ng/mL for the 1.3 mg/m² dose. The mean elimination half-life of bortezomib upon multiple dosing ranged from 40 to 193 hours. Bortezomib is eliminated more rapidly following the first dose. Mean Total Body Clearances were 102 and 112 L/h following the first dose for doses of 1.0 mg/m² and 1.3 mg/m², respectively, and ranged from 15 to 32 L/h following subsequent doses for doses of 1.0 and 1.3 mg/m², respectively. Clinical experience has shown that the change in clearance does not result in overt toxicity from accumulation in this multidose regimen in humans.

In subjects with advanced malignancies, the maximum pharmacodynamic effect (inhibition of 20S activity) occurred within 1-hour post dose. At the therapeutic dose of 1.3 mg/m² in subjects with multiple myeloma, the mean proteasome inhibition at 1-hour post dose was approximately 61%.

The time course of proteasome inhibition in subjects is characterized by maximum inhibition observed within the first hour after administration, followed by partial recovery of proteasome activity over the next 6 to 24 hours to within 50% of the pretreatment activity. On the Day 1, 4, 8, and 11 schedule, variable (10%–30%) levels of proteasome inhibition have been observed at next scheduled dosing. In theory, this advantage allows cells to recover proteasome activity for normal cellular housekeeping functions between doses.

The relationship between bortezomib plasma concentrations and proteasome inhibition can be described by a maximum effect ( $E_{max}$ ) model. The  $E_{max}$  curve is initially very steep, with small changes in plasma bortezomib concentration over the range of 0.5 to 2.0 ng/mL relating to large increases in the percent inhibition (0–60%). After that, a plateau occurs where marginal increases of proteasome inhibition are observed in spite of large changes in plasma bortezomib concentrations.

#### 1.3.5 Clinical Experience

It is estimated that more than 55,000 patients have been treated with bortezomib, including patients treated through Millennium-sponsored clinical trials, Investigator-Initiated Studies, the US NCI Cancer Therapy Evaluation Program (CTEP), and with commercially available drug. Bortezomib has been commercially available since 13 May 2003.

The overall goal of the Millennium phase 1 program was to determine the MTD and dose-limiting toxicity (DLT) of bortezomib in a number of therapeutic settings involving subjects with various advanced malignancies. In a Phase I trial in patients with refractory hematologic malignancies, the MTD for a twice weekly for 4 weeks of a 42 day cycle was 1.04 mg/m²/dose, with DLTs of thrombocytopenia, hyponatremia, hypokalemia, fatigue, and malaise (Orlowski et al., 2002). The toxicity was greatest during the third and fourth weeks of therapy. In the 3-week schedule of bortezomib monotherapy (4 doses, given on Days 1, 4, 8, and 11 of a 21-day treatment cycle), the DLT occurred at 1.56 mg/m²/dose (3 subjects with Grade 3 diarrhea and 1 with peripheral sensory neuropathy). Therefore, the MTD at this schedule was 1.3 mg/m²/dose. In a 35-day treatment cycle with 4 weekly doses of bortezomib monotherapy, the MTD was 1.6 mg/m²/dose and DLT included hypotension, tachycardia, diarrhea, and syncope.

In phase 1 clinical studies, anti-tumor activity was reported in subjects with NHL, multiple myeloma, Waldenström's Macroglobulinemia, squamous cell carcinoma of the nasopharynx, bronchoalveolar carcinoma of the lung, renal cell carcinoma, and prostate cancer.

The safety and efficacy of bortezomib in subjects with multiple myeloma were investigated in two phase 2 clinical studies, studies M34100-024 (subjects with first relapse) (Jagannath et al, 2004) and M34100-025 (subjects with second or greater relapse and refractory to their last prior therapy) (Richardson et al, 2003). In M34100-025, 202 heavily pre-treated subjects with refractory multiple myeloma after at least 2 previous treatments received bortezomib, 1.3 mg/m² on Days 1, 4, 8, and 11 of a 21-day treatment cycle. The European Group for Blood and Marrow Transplant (EBMT) response criteria, as described by Blade (Blade et al., 1998) were utilized to determine disease response. CRs were observed in 4% of subjects, with an additional 6% of patients meeting all criteria for CR but having a positive immunofixation test. PR or better was observed in 27% of subjects, and the overall response rate (CR, PR and minor response [MR] combined) was 35%. Seventy percent of subjects experienced stable disease or better.

The phase 3 study (M34101-039) (Richardson et al, 2005), also referred to as the APEX study, was designed to determine whether bortezomib provided benefit (time to progression [TTP], response rate, and survival) to patients with relapsed or refractory MM relative to treatment with high-dose dexamethasone. The study was also designed to determine the

safety and tolerability of bortezomib relative to high-dose dexamethasone, and whether treatment with bortezomib was associated with superior clinical benefit and quality of life relative to high-dose dexamethasone. A total of 669 patients were enrolled and 663 patients received study drug (bortezomib: 331; dexamethasone: 332). Patients randomized to bortezomib received 1.3 mg/m<sup>2</sup> I.V. push twice weekly on days 1, 4, 8, and 11 of a 3-week cycle for up to eight treatment cycles as induction therapy, followed by 1.3 mg/m<sup>2</sup> bortezomib weekly on days 1, 8, 15, and 22 of a 5-week cycle for three cycles as maintenance therapy. Patients randomized to dexamethasone received oral dexamethasone 40 mg once daily on days 1 to 4, 9 to 12, and 17 to 20 of a 5-week cycle for up to four treatment cycles as induction therapy, followed by dexamethasone 40 mg once daily on days 1 to 4 followed of a 4-week cycle for five cycles as maintenance therapy. The European Group for Blood and Marrow Transplant (EBMT) response criteria, as described by Blade (Blade et al., 1998) were utilized to determine disease response. There was a 78% increase in TTP for the bortezomib arm. Median TTP was 6.2 months for the bortezomib arm and 3.5 months for the dexamethasone arm (P<.0001). CR (complete response) + PR (partial response) was 38% with bortezomib vs. 18% with dexamethasone (P<.0001). CR was 6% with bortezomib vs. <1% with dexamethasone (P<.0001). The CR + nCR rate was13% with bortezomib vs. 2% with dexamethasone. In patients who had received only one prior line of treatment (bortezomib: 132; dexamethasone: 119), CR + PR was 45% with bortezomib vs. 26% with dexamethasone (P=.0035). With a median 8.3 months of follow-up, overall survival was significantly longer (P=.0013) for patients on the bortezomib arm vs. patients on the dexamethasone arm. The probability of survival at one year was 80% for the bortezomib arm vs. 66% for the dexamethasone arm, which represented a 41% decreased relative risk of death in the first year with bortezomib (P=.0005). In patients who had received only one prior line of treatment, the probability of survival at one year was 89% for the bortezomib arm vs. 72% for the dexamethasone arm, which represented a 61% decreased relative risk of death in the first year with bortezomib (P=.0098). (Richardson et al., 2005). Updated response rates and survival data were reported for M34101-039 (Richardson ASH, 2005). The updated CR (complete response) + PR (partial response) rate was 43% with bortezomib. The CR + nCR rate was 16% with bortezomib. With a median 22 months of follow-up, overall survival was significantly longer for patients on the bortezomib arm vs. patients on the dexamethasone arm. The median overall survival was 29.8 months (95% CI: 23.2, not estimable) for the VELCADE arm vs. 23.7 months (95% CI: 18.7, 29.1) for the dexamethasone arm (hazard ratio = 0.77, P= 0.0272). The probability of survival at one year was 80% for the bortezomib arm vs. 67% for the dexamethasone arm (P=0.0002).

Studies using bortezomib as monotherapy and in combination with other chemotherapy agents are continuing. Potential Risks of bortezomib (this section reflects updates to our

standard risks language that have been updated since I gave the modified version of the protocol several months ago.

#### 1.4 Combination of Bortezomib and Other Agents

A pre-clinical study reported by the Dana Farber Jerome Lipper Multiple Myeloma Center demonstrated synergy in cell line kill between bortezomib and other agents such as doxorubicin and melphalan (Mitsiades et al., 2003). Synergy was found with co-incubation of bortezomib with doxorubicin, or with pre-exposure to either of the drugs. Bortezomib exposure after prior doxorubicin exposure achieved the greatest cell kill. Myeloma cell lines known to be resistant to doxorubicin or melphalan confirmed sensitization by bortezomib, as did studies involving freshly isolated myeloma cells from patients known to be resistant to bortezomib or doxorubicin. A proposed mechanism for this enhancement of chemosensitivity is the down-regulation of several effectors involved in the cellular response to genotoxic stress, restoring sensitivity to DNA-damaging chemotherapeutic agents.

Berenson et al recently published a phase I/II trial of bortezomib and low-dose melphalan combination therapy for the treatment of patients with relapsed or refractory multiple myeloma (Berenson et al., 2006). Bortezomib was administered from 0.7 to 1.0 mg/m² on days 1, 4, 8, and 11 of a 28-day cycle for up to eight cycles, and oral melphalan was administered in escalating doses form 0.025 to 0.25 mg/kg on days 1 to 4. Thirty-five patients were enrolled and dose-limiting grade 4 neutropenia in two of six patients in the highest dose cohort led to the assignment of bortezomib 1.0 mg/m2 and melphalan 0.10 mg/kg as the maximum-tolerated dose. Responses were observed in 23 of 34 evaluable patients. Myelosuppression was the most prominent toxicity; Grade 1/2 neurotoxicity developed in 8 patients and worsened in 4 of 15 patients with pre-existing neurotoxicity. Diarrhea and nausea/vomiting were observed at all dose levels and no relationship to drug dosage was evident.

Hollmig et al. described treatment of 37 patients with bortezomib and high-dose melphalan (Hollmig et al., 2004). Bortezomib was dosed at 1.0 mg/m² or 1.3 mg/m² on days -4 and -1 before autologous HSC transplantation, with melphalan (50-200 mg/m²) given on the same days for 26 patients and on day -1 only for 11 patients. All patients achieved granulocyte (median, 13 days) and platelet (median, 17 days) recoveries. Serious (grade 3/4) mucositis and/or diarrhea occurred in 14% and 29% of patients, respectively. No transplant-related deaths were reported. A partial or better response was observed in 73% of evaluable patients. This same group also reported the use of 3 or 4 fractions of high-dose melphalan given along with bortezomib (1.0 or 1.3 mg/m²) in a standard day 1, 4, 7, ±10 fashion (Pineda-Roman et al., 2006). Maximum doses of melphalan reached 240-250 mg/m². Only 1 of 22 patients treated experienced significant (grade 2) mucositis with grade 3/4 diarrhea (primarily infectious) in 8 patients. These reports suggest a safe starting dose of bortezomib in combination with high-dose melphalan of 1.0 mg/m².

A similar phase I trial of bortezomib and pegulated liposomal doxorubicin (PegLD) enrolled 42 patients (24 with multiple myeloma) with advanced hematological malignancies (Orlowski et al., 2005). Bortezomib dosing started at 0.9 mg/m² and was advanced in a modified Fibonacci escalation with subsequent steps of 1.05, 1.2, 1.3, 1.4, and 1.5 mg/m², and was given on days 1, 4, 8, and 11 of each 21-day cycle. PegLD, 30 mg/m², was given on day 4 of each cycle. A bortezomib dose of 1.3 mg/m² was recommended for further study because of frequent dose reductions and delays at the MTD of 1.5 mg/m². Hematological toxicities were the most common, with fatigue being the most-common non-hematological toxicity. Again, diarrhea was observed at all dose levels. Of the 22 evaluable patients treated for myeloma, 8 achieved a CR or very good PR, and another 8 achieved a PR.

The combination of bortezomib and carboplatin was studied in a phase I trial involving 15 patients with recurrent ovarian or primary peritoneal cancer (Aghajanian et al., 2005). Carboplatin was administered on day 1 at a dose of 5 (AUC), and bortezomib on days 1, 4, 8, and 11 of each three week cycle at dose levels of 0.75, 1, 1.3, and 1.5 mg/m². No dose-limiting hematological toxicities were observed; dose-limiting non-hematological toxicities were diarrhea, skin rash, and sensory peripheral neuropathy (all grade 3) and the highest dose level of 1.5 mg/m², and the MTD was determined to be 1.3 mg/m². An overall response rate of 47% was demonstrated, and one patient with platinum-resistant disease achieved a CR.

We are conducting a phase I/II clinical study of bortezomib with dose-intense melphalan with autologous peripheral blood stem cell transplantation in patients with disease progression or less than partial response after a prior PBSCT (Rowley, et al, 2009). Primary exclusion criteria are active infection at time of PBSCT, cardiac amyloid deposition, and creatinine clearance of <20 ml/min. Peripheral neuropathy of less than grade 4 is not an exclusion. Bortezomib is given on days -4 and -1 with melphalan 200 mg/m² (actual weight) given on day -2 before PBSCT. For the phase I study, bortezomib was given at rising doses of 1.0, 1.3, and 1.6 mg/m². Three patients were to be enrolled at each dose level, with an additional 3 patients enrolled in case of a serious toxicity event at any level. An additional 20 patients are being enrolled in the phase II portion of the study with 15 patients enrolled as of 12/1/09 (patient accrual will be completed before enrollment into this study).

Twelve patients (median age, 58 yrs) were treated in the phase I study with 6 patients treated at the 1.0 mg/m² level after 1 patient experienced a serious adverse event (SAE) of prolonged diarrhea, and 3 patients treated at each of the subsequent levels. Eleven patients had 1 prior and 1 patient tandem prior cycles of dose-intense melphalan. All patients experienced the expected pancytopenia requiring red cell and/or platelet support. Ten

patients had febrile neutropenia with bacteremia identified in 3 patients. One patient had mild tumor lysis not requiring medical intervention. Mucositis was minimal and comparable to PBSCT with melphalan alone. All patients engrafted at a median time to ANC>500/uL of 11 days (range, 9-19) and platelet>20,000/uL of 14 days (range, 11-27). No other SAEs occurred in the phase I study beyond the usual events of high-dose therapy. No neurological SAEs, including severe peripheral neuropathies, were observed. A bortezomib dose of 1.6 mg/m² was chosen for the phase II study.

Fifteen patients (median age, 56 yrs) are now treated in the phase II study. Six patients had disease progression and 9 patients had less than a partial response (PR) after a prior PBSCT. All patients experienced pancytopenia and evaluable patients engrafted with median time to ANC>500/uL of 10 days (range, 8-13) and platelet>20,000 of 11 days (range, 9-65). Eleven patients had febrile neutropenia with 3 patients with positive blood cultures and 1 patient with RSV bronchitis. Three SAEs are reported in the phase II portion: 1 patient expired of complications of Candida krusei infection and 1 of MRSA sepsis (before ANC recovery). A third patient developed tumor lysis requiring dialysis. One patient had a dysphoric reaction to anti-emetics and did not receive the 2nd bortezomib dose. No neurological SAEs attributable to this regimen were observed in this population.

Patients underwent restaging studies at monthly intervals after transplantation with marrow examination at 3 and 12 months. Response classification is in accordance to standard definitions. Three patients underwent subsequent allogeneic PBSC and 2 patientss died of transplant-related complications and are not evaluable for response. Two patients succumbed to progressive disease. The remaining 20 patients are in ongoing follow-up. Eight patients including 6 of 11 patents with stable disease or minimal response after prior dose-intense melphalan achieved a CR. Six patients remain in continuous CR at 11+ to 23+ months (median, 15+ months) after PBSCT with 2 patients having disease progression at 12 and 26 months after PBSCT.

These data indicate that bortezomib can be added to dose-intense melphalan in this schedule with acceptable toxicities. Strikingly, 8 of 22 pts achieved CR after minimal response to dose-intense melphalan alone or disease progression after a prior PBSCT, and 2 patients showed tumor lysis, indicating a synergistic effect of adding bortezomib to dose-intense melphalan.

# 2 Study Objectives

# 2.1 Primary Objective:

To determine the progression-free survivals of patients with multiple myeloma treated with tandem cycles of high-dose melphalan followed by high-dose melphalan in combination with bortezomib with autologous HSC transplantation.

# 2.2 Secondary Objectives:

To determine the response rate, overall survival, and regimen-related toxicities of patients with multiple myeloma treated with high-dose melphalan or high-dose melphalan in combination with bortezomib given in tandem transplants

#### 3 Investigational Plan

#### 3.1 Overall Design and Plan of Study

This is a multi-institution phase II non- randomized study

#### 3.2 Patient Selection

- 3.3 Inclusion Criteria (1st and 2nd transplants)
  - 3.3.1 Confirmed diagnosis of multiple myeloma with either a
    Durie-Salmon stage I, II, or III or ISS stage I, II or III, less than 12
    months since initiation of systemic therapy
  - 3.3.2  $\geq 8x10^6$  CD34+cells/kg available in cryopreservation in aliquots

appropriate for tandem transplants

- 3.3.3 Age: 18-75 years at time of transplantation
- 3.3.4 KPS 70-100%
- 3.3.5 Recovery from complications of prior therapies
- 3.3.6 Gender: There is no gender restriction

# 3.4 Exclusion Criteria (1st and 2nd transplants)

Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

- 3.4.1 Diagnosis other than multiple myeloma
- 3.4.2 Chemotherapy or radiotherapy within 8 days of initiating treatment in this study
- 3.4.3 Prior autologous or allogeneic transplantation (except as enrolled into this study)
- 3.4.4 Uncontrolled bacterial, viral, fungal or parasitic infections
- 3.4.5 Uncontrolled CNS metastases
- 3.4.6 Known amyloid deposition in heart
- 3.4.7 Organ dysfunction
  - 3.4.7.1 LVEF <40% or cardiac failure not responsive to therapy
  - 3.4.7.2 FVC, FEV<sub>1</sub>, or DLCO <40% of predicted and/or receiving supplementary continuous oxygen

- 3.4.7.3 Evidence of hepatic synthetic dysfunction, or total bilirubin >2x or AST >3x ULN
- 3.4.7.4 Calculated creatinine clearance <20 ml/min
- 3.4.8 Sensory peripheral neuropathy grade 4 within 14 days of enrollment
- 3.4.9 Karnofsky score <70% unless a result of bone disease directly caused by myeloma
- 3.4.10 Life expectancy limited by another co-morbid illness
- 3.4.11 Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
- 3.4.12 Female subject is pregnant or breast-feeding (women) or unwilling to use acceptable birth control methods (men or women) for twelve months after treatment. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
- 3.4.13 Documented hypersensitivity to melphalan or to bortezomib, boron or mannitol or any components of the formulation
- 3.4.14 Patients unable or unwilling to provide consent
- 3.4.15 Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant
- 3.4.16 Patient has received other investigational drugs with 14 days before enrollment
- 3.4.17 Serious medical or psychiatric illness likely to interfere with participation in this clinical study

# 3.5 Patient Evaluations – First Transplant

- 3.5.1 Pre-transplant evaluation must be performed within 60 days of transplant, except for HLA, ABO and Rh typing
- 3.5.2 History with full details of the patient's prior treatments and responses
- **3.5.3** Careful physical exam with determination of Karnofsky score and findings related to underlying malignancy
- 3.5.4 Chemistry profile to include serum creatinine, AST, alkaline phosphatase, and bilirubin
- 3.5.5 CBC with differential
- 3.5.6 ABO, Rh, red cell antibody screen
- 3.5.7 PT, PTT
- 3.5.8 Serum pregnancy test, if female gender with child-bearing potential
- 3.5.9 HIV, Hepatitis B, Hepatitis C and CMV serology
  - 3.5.9.1 Infectious disease testing, if previously documented positive, need not be repeated to comply with this requirement.
- 3.5.10 Creatinine clearance (calculated)
- 3.5.11 Disease Staging
  - 3.5.11.1 Serum and urine protein electrophoreses and immunofixation with measurement of monoclonal protein
  - 3.5.11.2 **B2M**
- 3.5.12 Radiological studies of any sites of bone pain or bone scan abnormalities
- 3.5.13 Skeletal survey if not performed within 6 months of start of study treatment
- 3.5.14 Pulmonary function tests with DLCO
- 3.5.15 MUGA scan or cardiac echo

3.5.16 Patients with a suspected diagnosis of amyloidosis will undergo echocardiography for the detection of cardiac involvement

#### 3.5.17 EKG

# 3.6 Patient Evaluations – Second Transplant

- **3.6.1** History with full details of the patient's prior treatments and responses
- 3.6.2 Careful physical exam with determination of Karnofsky score and findings related to underlying malignancy
- 3.6.3 Chemistry profile to include serum creatinine, AST, alkaline phosphatase, and bilirubin
- 3.6.4 CBC with differential
- 3.6.5 ABO, Rh, red cell antibody screen
- 3.6.6 PT, PTT
- 3.6.7 Serum pregnancy test, if female gender with child-bearing potential
- 3.6.8 HIV, Hepatitis B, Hepatitis C and CMV serology
  - 3.6.8.1 Infectious disease testing, if previously documented positive, need not be repeated to comply with this requirement.
- 3.6.9 Creatinine clearance (calculated)
- 3.6.10 Disease Staging
  - 3.6.10.1 Serum and urine protein electrophoreses and immunofixation with measurement of monoclonal protein
  - 3.6.10.2 β2m
  - **3.6.10.3** Radiological studies of any sites of bone pain or bone scan abnormalities

#### 3.7 Analysis of PBSC and Marrow Components

**3.7.1** TNC and CD34+ cell count

#### 3.8 Post-Transplant Evaluation

- **3.8.1** Physical exam, daily until hematological recovery and resolution of serious regimen-related complications
- 3.8.2 Daily assessment of toxicity from day-1 until resolution of all Grade 3/4 treatment-related toxicities
  - 3.8.2.1 Presence assessed and scored in accordance with NCI toxicity guidelines
- 3.8.3 CBC daily from day 0 until ANC ≥500/ul on two sequential days after nadir reached (engraftment). Thereafter, CBC at least weekly until documentation of transfusion independence (platelet count ≥20,000/ul without transfusion for ≥7 days)
- 3.8.4 Chemistry profile including magnesium t.i.w. until documentation of engraftment, and then at least weekly until stabilization of electrolytes is documented
- 3.8.5 Record of all medications administered during inpatient course

#### 3.9 Post transplant re-staging of disease

- 3.9.1 Restaging by serum and urine should be done at 4 weeks intervals (±7 days) starting at day +28 after transplantation for 3 months and then at 3 months intervals until 3 years after transplantation or demonstration of disease progression requiring therapy, if earlier.
- **3.9.1.1** Staging studies will be obtained after both 1<sup>st</sup> and 2<sup>nd</sup> transplants.
- 3.9.2 24 hour urine for creatinine clearance, total protein, protein electrophoresis with quantitation of monoclonal protein by immunofixation, serum free light chain measurements at 4 week intervals (±7 days) starting at day +28 after transplantation for 3 months and then at 3 month intervals (or more frequently as clinically necessary) until demonstration of disease progression

3.9.2.1 Staging studies will be obtained after both 1<sup>st</sup> and 2<sup>nd</sup> transplants.

#### 3.10 Study Treatments

# 3.10.1 Study Medications

3.10.1.1 Bortezomib (VELCADE) for Injection is a sterile lyophilized powder for reconstitution and is supplied in vials containing bortezomib and mannitol at a 1:10 ratio. For example, vials containing 3.5 mg of bortezomib contain 35 mg of mannitol. Vials containing lyophilized bortezomib for Injection should be stored according to the label requirements. For the United States, store at USP Controlled Room Temperature which is 25°C (77°F); excursions permitted from 15 to 30°C (59 to 86°F). For Europe, do not store above 30°C (86°F). To date, stability data indicate that the lyophilized drug product is stable for at least 18 months when stored under the recommended conditions. Stability studies are ongoing, and Millennium Pharmaceuticals, Inc. will notify the investigator should this information be revised during the conduct of the study. bortezomib is cytotoxic. As with all cytotoxic drugs, caution is required when preparing and handling bortezomib solutions. Cytotoxic drugs should only be handled by staff specially trained in the safe handling of such preparations. The use of gloves and other appropriate protective clothing is recommended. In case of skin contact, wash the affected area immediately and thoroughly with soap and water for at least 15 minutes. If product contacts eye, immediately flush eye thoroughly with water for at least 15 minutes. Always contact a physician after any form of body contact. All materials that have been used for preparation should be disposed of according to standard practices. A log must be kept of all disposed materials. The drug is available in sterile, single use vials containing 3.5 mg of bortezomib. Each vial of bortezomib for Injection should be reconstituted under a laminar flow biological cabinet

(hood) within eight hours before dosing with 3.5 mL of normal (0.9%) saline, Sodium Chloride Injection USP, so that the reconstituted solution contains bortezomib at a concentration of 1 mg/mL. Prior to reconstitution the vials should remain in the cartons to protect them from light. Dissolution is completed in approximately 10 seconds. The reconstituted solution is clear and colorless, with a final pH of 5 to 6. Reconstituted bortezomib should be administered promptly and in no case more than 8 hours after reconstitution. All materials that have been used for preparation should be disposed of according to standard practices. A log must be kept of all disposed material.

3.10.1.2

Melphalan for Injection is a sterile lyophilized powder for reconstitution and will be obtained from the manufacturer in accordance with standard pharmacy purchasing criteria. Melphalan will be reconstituted by pharmacy staff, in accordance with usual pharmacy practices, immediately before patient infusion. Melphalan is a bifunctional alkylating agent that acts principally through covalent reactions with DNA, resulting in the formation of drug-DNA adducts with cross-linking of DNA strands. Melphalan's cytotoxic effects are related to its concentration and the duration of exposure to melphalan of the cell. Enhanced repair of DNA interstrand crosslinks may be a mechanism of resistance that develops after prior exposure to this drug. Melphalan is actively transported into cells by the high-affinity L-amino acid transport system; glutamine and leucine compete for carrier uptake and high levels of these amino acids can reduce drug uptake. Other drugs such as tamoxifen, chlorpromazine, and indomethacin can also impair melphalan uptake and accumulation. Studies of the pharmacokinetics of oral melphalan were complicated by the highly variable absorption of the drug. Moreover, studies of intravenous melphalan have also showed considerable inter-patient variability in plasma clearance.

Pinguet et al studied the pharmacokinetics of melphalan administered at a dose of 140 mg/m<sup>2</sup> in combination with other chemotherapeutic agents to 20 patients undergoing autologous PBSC transplantation. The medians time to neutrophil and platelet recoveries were 16 and 14.6 days, and the majority of patients (80%) developed WHO grade 3/4 stomatitis. Plasma concentration profiles were biphasic and fitted with a two-compartment model. The maximal concentration at the end of infusion averaged  $7.94\pm3.73$  mg/l (range, 1.65-14.5). The mean elimination half-life and the mean residence time were 83.1±27.1 minutes (range, 51.6-166.81) and 98.7±26.9 minutes (range 59.5-166.9), respectively. The volume of distribution averaged 1.00±0.62 l/kg (range 0.46-3.12) and total plasma clearance 548.3±300.0 ml/min/m<sup>2</sup> (range, 218.6-1378.8). Plasma levels were below the limits of detection for all patients by 24 hours after melphalan administration. These authors noted large inter-individual variability of these pharmacokinetic parameters. Total clearance of melphalan was significantly correlated with creatinine clearance (r=0.49, p<0.05). A relationship between melphalan clearance and renal function was also described by Kergueris et al., but this relationship did not explain the large variation in inter-individual overall clearance of the drug (Kergueris et al., 1994). Similar pharmacokinetic results were reported for 20 pediatric and 10 adult patients treated with melphalan 140 mg/m<sup>2</sup> as a single agent. For the adult patients, the elimination half-life ( $t^{1/2}\beta$ ) was  $50\pm7$  minutes for patients treated with  $140 \text{ mg/m}^2$  dose and  $41\pm12$ minutes for the higher dose of 180 mg/m<sup>2</sup>. Plasma clearance averaged 525 ml/min/m<sup>2</sup> at 140 mg/m<sup>2</sup> and 532  $ml/min/m^2$  at 180  $mg/m^2$ .

#### 3.11 Outline of Treatment Plan

Patients will sequentially undergo two transplants in this order.

Figure 1: Outline of Treatment Schema First Transplant

 $\begin{array}{c} \text{Melphalan 200 mg/m2 day -1} \\ & \downarrow \\ \text{Autologous HSCT} \end{array}$ 

Figure 2: Outline of Treatment Schema Second Transplant

Bortezomib 1.6 mg/m2 d-4

Welphalan 200mg/m2 d-2

Bortezomib 1.6mg/m2 d-1

Autologous HSCT

#### 3.12 Conditioning Regimens

- 3.12.1 First Transplant
- 3.12.2 Melphalan
  - 3.12.2.1 Melphalan is administered by rapid intravenous infusion via a central vein over one hour
  - 3.12.2.2 The final dilution of melphalan is physically and chemically stable for 60 minutes and therefore will be administered within that time period
  - 3.12.2.3 Melphalan will be given as a single dose (not split over 2 or more days)
  - 3.12.2.4 Patients are encouraged to "chew" ice for 15 minutes before through 1 hour after administration of melphalan
  - 3.12.2.5 Dosing will be based on body surface area calculated using actual body weight
  - 3.12.2.6 Patients will be hospitalized starting at least 1 hr before melphalan administration and continuing for at least 10 days after melphalan infusion (may be discharged home on day +10). Aggressive hydration will be used for uro-protection during the time of melphalan administration and for 24 hours after the completion of melphalan infusion

#### 3.13 Second Transplant

#### 3 14 Bortezomib

- 3.14.1 Bortezomib is administered by rapid I.V. push (over 3-5 seconds) via a central or peripheral vein into a flowing saline line
- 3.14.2 Bortezomib will be administered any time on day -4, at least 20 hrs after the start of the melphalan infusion on day -1
- 3.14.3 Dosing will be based on body surface area calculated using actual body weight

3.14.4 Dexamethasone is administered at a dose of 20 mg i.v. daily on days -4 and -1 (with bortezomib). Dexamethasone is administered at a dose of 10 mg i.v. as a component of the anti-nausea regimen on day -2 before melphalan administration

#### 3.15 Stem Cell Infusion

- 3.15.1 Day 0 is defined as the day of first stem cell infusion.
- 3.15.2 Additional cells may be infused on subsequent days if the volume of the HSC components is deemed too large for a single infusion
- 3.15.3 HSC will be infused at least 18 hrs or later after bortezomib infusion
- 3.15.4 Day 0 should be fixed on a Monday Friday, when possible
- 3.15.5 All patients will receive unmodified HSCT (other than cryopreservation). These components will not be irradiated
- 3.15.6 Cells will be infused according to HUMC Standard Practice guidelines

#### 3.16 Post-transplant Cytokine Administration.

3.16.1 Patients will routinely receive filgrastim, 5 ug/kg sc, on days 3, 5, 7, 9 and 10+ after stem cell transplantation. Filgrastim dose may be rounded to vial size (e.g., <70kg: 300 ug, 70-90 kg: 480 ug, >90 kg: 600 ug)

#### 3.17 Post-transplant Supportive Care

**3.17.1** Hospitalization: Patients will cared for in the inpatient or outpatient transplant units. Patients will be discharged from the transplant unit when hematological recovery occurs, the patient is clinically stable, and all grade 3/4 toxicities have resolved, but not before day +10 of transplantation

#### 3.17.2 Mucositis

Patients may receive any anti-emetic regimen determined to be clinically appropriate

- **3.17.2.2** Patients may receive any anti-diarrhea regimen determined to be clinically appropriat
- 3.17.3 Central line: Patients will have central venous access suitable for TPN and blood component support and maintained according to HUMC Standard Practice guidelines
- 3.17.4 Infection prophylaxis: Patients will receive prophylaxis for PCP, HSV, bacterial, and fungal infections according to HUMC Standard Practice guidelines
- 3.17.5 Blood component support: Patients will receive transfusions in accordance with HUMC Standard Practice guidelines
- 3.17.6 Nutrition: Patients may receive enteral or parenteral alimentation if caloric or protein intake falls below daily basal needs
- 3.17.7 Post-transplant treatment: There are no restrictions for administration of involved field radiation, chemotherapy, maintenance therapy, or surgical interventions after transplantation
- 3.17.8 Bisphosphinates: Monthly infusions of bisphosphinate therapy after transplantation should be considered for all patients
- 3.17.9 Post-transplant vaccinations: Vaccinations will be administered after transplantation in accordance with HUMC Standard Practice guidelines

#### 3.18 Disease Response

**3.18.1** Patients should undergo restaging of disease at 4 week intervals starting one month after transplant as defined in section 3.9

#### 3.19 Timing between Transplant Procedures

Patients will undergo  $2^{nd}$  transplant (day 0) no earlier than day 84 and no later than day 180 after the  $1^{st}$  transplant (day 0)

#### 3.20 Dosing of Agents

**3.20.1** Melphalan dosing will be based on actual body weight. The amount (in mg) of drug to be administered will be determined

- based on body surface area. Body surface area is to be calculated based on body weight using a standard nomograM
- 3.20.2 Bortezomib dosing will be based on actual body weight. The amount (in mg) of drug to be administered will be determined based on body surface area. Body surface area is to be calculated based on body weight using a standard nomogram
- 3.20.3 Patient weight will be determined by the nursing or nutrition staff within 7 days of start of conditioning
- 3.20.4 Administration of Melphalan
  - 3.20.4.1 Melphalan will be dosed based on actual body weight at a dose of 200 mg/m² and infused on day -1 (first transplant) or day -2 (second transplant)
  - 3.20.4.2 Administer melphalan IV over one hour through a central catheter. Rapid infusion may result in dizziness, nasal stuffiness, rhinorrhea, or nasal congestion during or immediately after infusion
  - 3.20.4.3 Administer early in the day
  - 3.20.4.4 Have patient empty bladder frequently
  - 3.20.4.5 Patients will receive hydration before and after administration of melphalan
  - 3.20.4.6 "Chewing" on ice may decrease the severity of oral mucositis and is encouraged for all patients starting 15 minutes before, during, and for 60 minutes after the infusion of melphalan
  - 3.20.4.7 Patients will receive an anti-emetic regimen of dexamethasone 10 mg i.v., and ondansetron 12 mg i.v. 30 minutes before melphalan infusion
- 3.20.5 Administration of Bortezomib
  - 3.20.5.1 Bortezomib will be dosed based on actual body weight and infused on day -4, and day -1 before HSC infusion
  - 3.20.5.2 Bortezomib is supplied as a lyophilized white powder in 3.5 mg single-dose vials

- 3.20.5.3 Bortezomib is reconstituted with 1.2 ml sterile water for injection, without shaking
- 3.20.5.4 Administration
  - 3.20.5.4.1 Rapid I.V. push over 3-5 seconds via a central or peripheral vein. Each vial is for a single use administration.
  - 3.20.5.4.2 Second dose of bortezomib will be no less than 20hrs after melphalan administration
  - 3.20.5.4.3 Dexamethasone, 20 mg i.v., will be given as a pre-medication.

#### 3.21 Pre-Transplant Therapy

Chemotherapy and/or radiation therapy may be given to reduce tumor bulk as determined on clinical grounds. The referring oncologist may be asked to administer this therapy. The prior therapies are not specified by this protocol

- 3.21.1 Patients will not proceed to dose-intense therapy any sooner than 8 days after completion of the most recent cycle of chemotherapy or radiotherapy
  - 3.21.1.1 The timing of therapy is in reference to the dose of melphalan
  - 3.21.1.2 Therapy with thalidomide and/or corticosteroids may be discontinued no less than 7 days before initiation of bortezomib
- 3.21.2 Collection of Autologous Hematopoietic Stem Cells

The methods of collection of hematopoietic stem cells are not specified by this protocol

#### 3.22 Treatment Assignment

All patients will undergo the same treatment regimen

#### 3.23 Blinding, Packaging, and Labeling

VELCADE will be supplied in vials as open-label stock. Both the box label and vial label will fulfill all requirements specified by governing regulations.

Melphalan will be supplied in vials as open-label stock. Both the box label and vial label will fulfill all requirements specified by governing regulations.

#### 3.24 Concomitant Treatment

3.24.1 Required Concurrent Therapy

Not applicable. Patients will receive standard care

3.24.2 Prohibited Concurrent Therapy

Any investigational agent

### 3.25 Treatment Compliance

All drug will be administered to eligible patients under the supervision of the investigator or identified sub-investigator(s). The pharmacist will maintain records of drug receipt (if applicable), drug preparation, and dispensing, including the applicable lot numbers, patients' height, body weight, and body surface area, and total drug administered in milliliters and milligrams. Any discrepancy between the calculated dose and dose administered and the reason for the discrepancy must be recorded in the source documents

# 3.26 Duration of Treatment and Patient Participation

Patients will be hospitalized until at least day +10 after transplantation and resolution of serious adverse events. Patients will then be followed, indefinitely, for survival and duration of response to the treatment received.

#### 3.27 Termination of Treatment and/or Study Participation

Patients will be informed that they have the right to withdraw from the study at any time for any reason, without prejudice to their medical care. The investigator also has the right to withdraw patients from the study for any of the following reasons:

- Intercurrent illness
- Occurrence of an unacceptable adverse event
- Patient request
- Protocol violations
- Non-compliance
- Administrative reasons
- Failure to return for follow-up

- General or specific changes in the patient's condition unacceptable for further treatment in the judgment of the investigator
- Progressive disease at any time

At the time of withdrawal, all study procedures outlined for the End of Study visit should be completed. The primary reason for a patient's withdrawal from the study is to be recorded in the source documents.
#### 4 Adverse Events

#### 4.1 Definitions

#### 4.1.1 Adverse Event Definition

An adverse event (AE) is any untoward medical occurrence in a patient administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. An adverse event can be any unfavorable and unintended sign (eg, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the drug, whether or not it is considered to be drug related. This includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of drug.

#### 4.1.2 Serious Adverse Event Definition

A serious adverse event (SAE) is any adverse event, occurring at any dose and regardless of causality that:

- Results in death.
- Is life-threatening. Life-threatening means that the patient was at immediate risk of death from the reaction as it occurred, i.e., it does not include a reaction which hypothetically might have caused death had it occurred in a more severe form.
- Requires inpatient hospitalization or prolongation of existing hospitalization.
  Hospitalization admissions and/or surgical operations scheduled to occur during the
  study period, but planned prior to study entry are not considered AEs if the illness or
  disease existed before the patient was enrolled in the trial, provided that it did not
  deteriorate in an unexpected manner during the trial (eg, surgery performed earlier than
  planned).
- Results in persistent or significant disability/incapacity. Disability is defined as a substantial disruption of a persons' ability to conduct normal life functions.
- Is a congenital anomaly/birth defect.
- Is an important medical event. An important medical event is an event that may not result in death, be life-threatening, or require hospitalization but may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the definitions for SAEs. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

Clarification should be made between the terms "serious" and "severe" since they ARE NOT synonymous. The term "severe" is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as a severe headache). This is NOT the same as "serious," which is based on patient/event outcome or action criteria described above and are usually associated with events that pose a threat to a patient's life or functioning. A severe adverse event does not necessarily need to be considered serious. For example, persistent nausea of several hours duration may be considered severe nausea but not an SAE. On the other hand, a stroke resulting in only a minor degree of disability may be considered mild, but would be defined as an SAE based on the above noted criteria. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

# 4.2 Procedures for AE and SAE Reporting

Investigator-sponsor must report all serious adverse event (SAE) regardless of relationship with any study drug or expectedness to the IRB as required by the institution.

Intensity for each adverse event, including any lab abnormality, will be determined by using the NCI CTCAE, version 3.0, as a guideline, wherever possible. The criteria are available online at <a href="http://ctep.cancer.gov/reporting/ctc.html">http://ctep.cancer.gov/reporting/ctc.html</a>.

## 4.3 Assessment of Toxicity

- 4.3.1. Common Terminology Criteria for Adverse Events (CTCAE) will be used for the assessment and grading of all toxicities experienced by patients enrolled into this study (htt;:///ctep.cancer.gov/forms/CTCAE Index.pdf).
  - a. If the nature of the adverse experience is listed in the CTCAE, the maximum grade and time of maximum grade will be reported.
  - b. If the adverse experience is not listed on the NCI CTG Expanded Toxicity Criteria Appendix D, report the toxicity grade using the following criteria:
    - Grade 1= Mild: an adverse experience which is easily tolerated by the patient, causing minimal discomfort and not interfering with everyday activities.
    - Grade 2 = Moderate: an adverse experience which is sufficienty discomforting to interfere with normal every day activities.
    - Grade 3 = Severe: an adverse experience which is incapacitating and prevents normal every day activities.
    - Grade 4 = Life Threatening: an adverse experience which places the patient at immediate risk of death.

#### 4.3.2. Assessment of Causality

a. Every effort should be made by the investigator to explain each adverse experience and assess its relationship, if any, to study drug treatment.
 Causality should be assessed using the following categories: Not Related, Unlikely, Suspected (Reasonable Possibility), Probable.

Not related: The adverse experience is definitely not related to the test drug.

Unlikely: There are other, more likely causes and the drug is not suspected as a cause.

Suspected (reasonable possibility): A direct cause and effect relationship between the drug and the adverse experience has not been demonstrated but there is a reasonable possibility that the experience was caused by the drug.

Probable: There probably is a direct cause and effect relationship between the adverse experience and the study drug.

b. The degree of certainty with which an adverse experience is attributed to drug treatment (or alternative causes, e.g.: natural history of the underlying diseases, concomitant therapy, etc.) will be determined by how well the experience can be understood in terms of one or more of the following.

Known pharmacology of the drug

Reaction of similar nature being previously observed with this drug or class of drug. The experience having often been reported in literature for similar drugs as drug related e.g.: skin rashes, blood dyscrasia. The experience being related by time to drug ingestion terminating with drug withdrawal (dechallenge) or reproduced on rechallenge.

#### 4.3.3. Follow-up of Adverse Experiences

- a. Patients with adverse experiences will be actively followed until the event has subsided (disappeared) or until the condition has stabilized.
- b. Adverse events, both serious and non-serious, and deaths that occur during the patient's study participation will be recorded in the source documents. All SAEs should be monitored until they are resolved or are clearly determined to be due to a patient's stable or chronic condition or intercurrent illness(es).

#### 5 Statistical Evaluation

This is a phase II study to determine the progression-free survivals of patients with multiple myeloma treated with tandem cycles of high-dose melphalan followed by high-dose melphalan in combination with bortezomib with autologous HSC transplantation.

# 5.1 **Endpoint**

- 5.1.1 Primary Objective
  - 5.1.1.1 The main primary endpoint of this study is three-year progression free survival. Patients are considered a failure with respect to PFS if they die or experience disease progression or relapse. The time to this event is the time from transplantation to relapse/progression, initiation of non-protocol anti-myeloma therapy, or death from any cause. Subjects alive without confirmed disease progression will be censored at the time of last disease evaluation. Deaths without progression are treated as failures no matter when they occur.
- 5.1.2 Secondary Objective
- 5.2 5.2.1.1 To determine the response rate, overall survival, and regimen-related toxicities of patients with multiple myeloma treated with high-dose melphalan in combination with bortezomib given in tandem transplants

#### 5.2 Secondary endpoints will include:

- a. Overall response rates: Defined as the composite endpoint of response to treatment which includes Complete Response (CR), Partial Response (PR), stable disease (SD) as defined in International Response Criteria. We will also analyze Complete Response rate.
- b. Overall survival (OS): Defined as time from the first dose of administration to death from any cause.
- c. Univariate analysis of risk of progression/relapse and mortality: To examine the univariate effects of the prognostic features on the outcomes EFS and OS for patients using this modality with respect to risk of relapse/progression and death from any cause.
- d. Univariate analysis of the risk of progression/relapse and mortality: In addition, multivariate analysis of the risk of progression/relapse and overall mortality will be conducted to assess influence of variables measured after the start of treatment.
- e. Regimen-related toxicity: Graded and presented in a descriptive nature.

Descriptive analysis of baseline characteristics and demographics in this study will be performed in the following manner. Continuous measurements will be summarized as mean (SD) or median (inter-quartile range) based on whether or not the data come from a normal distribution as validated by Shapiro-Wilks test of normality. Categorical measurements will be summarized as frequency (percentage). Proportion of overall survival will be estimated by the Kaplan-Meier product limit method. The univariate probability of the relapse and treatment–related mortality (TRM) will be calculated using cumulative incidence function.

## 5.3 Accrual, Registration and Follow-up

The targeted sample size for the single arm is 97 subjects that successfully undergo the 2<sup>nd</sup> transplant. It is estimated that eight years 1 month (97 months) of accrual will be necessary to enroll this number of subjects. The Blood and Marrow Transplantation Program at HUMC treats over 120 patients with this diagnosis every year. In the last two years, an estimated 50 multiple myeloma patients each year underwent tandem autologous hematopoietic stem cell transplantation using the high-dose melphalan conditioning regimen. It is assumed that patients will enroll into the study uniformly over the accrual period at the rate 1 patient per month. After eligibility is established, subjects will be enrolled into the single arm using high-dose melphalan and high-dose melphalan-bortezomib as a conditioning regimen.

All subjects will be "on-study" for three years post-transplant, during which they will be monitored for the effects of treatment through regular clinic. With four years of planned accrual, and a minimum of three years of additional follow-up post-transplant, subjects will be followed for progression-free survival for at least 36 months.

# 5.4 Sample Size and Power Calculations

In this section, the power of the analysis of time to progression or death is considered and performed based on the proportion surviving without progression at three years. The standard tandem autologous HSCT with high-dose melphalan conditioning regimen is assumed to have PFS of 56%. It is posited that the high-dose melphalan and melphalan-bortezomib conditioning regimen will increase the three-year PFS to 76%. To estimate the 3-year PFS in tandem autologous HSCT followed by high dose Mel-Vel based on an anticipated advantage over 3-PFS observed in historical controls, the method of Simon and Dixon (9) was used to derive the sample size. At the design stage, it was stated that there were 150 patients in the historical control cohort who had received tandem auto HSCT with HD melphalan. Median event-free survival in the 150 was 3.58 years (42.96 months) and 44%(66 of 150) had had progression of disease. Hazard rate in the HC is 0.44 and hazard rate in the experimental arm (with melphalan-bortezomib) is 0.24 thus the ratio of the hazard rates is 1.8333. However, to adjust for the dropout due to MD decision, Patient decision, PD before 2<sup>nd</sup> transplant, or loss of insurance averaging to a rate 0.3, the hazard rate is (.44+.3)/(.24+.3)=1.37. If we assume accrual rate of 1 patient per month, 5% level of significance and 80%, a sample of 97 patients that successfully undergo the 2<sup>nd</sup> transplant will be required and this calculation will achieve 80.17% power to show that PFS is at least 76% in the single arm. Adjusted Sample Size

This is adjustment was not preplanned, however, after observing the slower accrual of 1 patient per month and the larger than anticipated dropouts post-first transplant, it was deemed necessary to employ an adjustment with respect to dropout, for the single arm versus historical control if the power to detect the efficacy of high-dose melphalan and high-dose melphalan-bortezomib were to be preserved.

#### 5.5 Efficacy analysis

This is a phase II study comparing the progression-free survival after tandem autologous HSCT with high-dose melphalan to high-dose melphalan and bortezomib in patients with a diagnosis of multiple myeloma.

# 5.6 Statistical Hypothesis

The null hypothesis is that the three-year progression free survival rate in multiple myeloma patients receiving tandem autologous HSCT with high-dose melphalan (control arm) is 56%. The alternative hypothesis for this study posits that the treatment plan consisting of tandem autologous HSCT with high-dose melphalan followed by high-dose melphalan-bortezomib (experimental arm) will increase the 3 year progression free survival to 76%, which is 20 % more than PFS in the historical arm. Note that the hazard rate for progression in historical tandem cohort,  $\lambda_c$ , is 0.44 (1-0.56) and the experimental arm with HD Mel-Vel has a hazard rate,  $\lambda_E$ , of 0.24 (1-0.76), so that the minimum hazard ratio,  $\delta = \lambda_c / \lambda_E$ , is 0.44/0.24=1.833. Thus this single arm trial of increased PFS at 3 years post-HSCT is equivalent to evaluating

hypotheses:

 $H_0$ : δ (3)≤1

 $H_A: \delta(3) > 1 S_E(3)$ 

where  $\delta$  (3) = the three-year progression of disease hazard ratio Thus, a one-sided log-rank test stratified on risk status will be conducted to determine if tandem autologous HSCT with high-dose melphalan and melphalan-bortezomib improves the progression free survival over that in historical controls using high-dose mephalan alone using a 5% level of significance. Equivalently, estimating a 90% confidence interval of the 3 year progression-free survival would achieve the desired goal.

#### 5.7 Primary endpoint

The primary analysis will include all eligible autologous transplantation subjects that receive the high-dose Mel-MelVel conditioning regimen and historical control of standard tandem HSCT recipients using high-dose melphalan conditioning regimen. 3 –year PFS and corresponding 90% confidence interval will be estimated using Kaplan-Meier method. It is anticipated that the estimated 90% confidence interval should include 76% and exclude 56% to show evidence that tandem autologous HSCT with high-dose melphalan and melphalan-bortezomib improves the progression-free survival in this patient population.

# 5.8 Secondary endpoints

## **5.8.1** Response to Treatment

The rates of complete remission (CR), and very good partial remission (VGPR) according to the International Uniform Response Criteria (Section 3.2) will be calculated at two years after transplantation. The analyses of the two-year response rates are planned as soon as those data become available in all subjects, at one and two years after the close of accrual. Estimated proportions or response and their corresponding exact binomial 95% confidence interval will be

reported for these endpoints. Fisher's exact test will be used to compare response to treatment for both CR and VGPR endpoints between any groups using 5% level of significance.

#### 5.8.2 Overall Survival

The event is death from any cause. The time to this event is the time from transplantation to death, loss to follow-up or the end of the study, whichever comes first. Patients alive at the time of last observation are considered censored. The Kaplan-Meier estimate of survival, along with corresponding with 90% confidence interval, will be computed at 1 year, 2 year and 3 year post tandem transplant for all patients and separately for any group. For any group comparisons, a log-rank test, conducted at a one-sided significance level of 0.05.

## 5.8.3 Association between Prognostic factors and EFS and OS

Ananalysis of risk outcomes relapse/progression, transplant-related mortality, and overall mortality will be conducted while adjusting for imbalance in other risk factors using a Cox proportional hazards model (10). To fit the multivariate model, a stepwise backward selection procedure will be used while considering relapse risk status (low risk, high risk), age at transplant and Karnosfky performance score (<90 versus ≥90). An examination of the goodness-of-fit will be performed using Grambsch-Therneau and Martingale residual plots (11) and Loess smooth of Cleveland (12). Covariates yielding a p-value of 0.05 or less will be an indication of statistical significance. The proportionality assumption for Cox regression will be validated by introducing a time-dependent covariate for each risk factor and outcome. This analysis will be presented in terms of relative risks (RR) along with the corresponding p values for each covariate.

## 5.9 Safety Analysis

Safety Analysis will be performed on all patients who have at least one dose of medication on either treatment arms over the course of this study. The severity of the toxicities will be graded according to the NCI CTCAE v3.0 whenever possible. Events during the first 100 days after transplantation will be considered possibly related to the transplant for this analysis. Regimen-related toxicity will be graded and presented in a descriptive nature as incidence rates and corresponding exact binomial 95% confidence intervals.

## 5.9.1 Safety Monitoring Endpoints

The incidence of toxicities of grade 3 or higher toxicities (CTCAE version 3.0), the incidence of probable viral fungal and bacterial infections, and the incidence of treatment-related morality, i.e., from causes other than relapse or progression, will be recorded for each patient at set intervals over the course of the study. Safety data will be described in a variety of ways, both graphical and tabular, and incidence will be compared across time points and treatment arms. The Data and Safety Monitoring Board will be presented with a comprehensive semi-annual report that will contain both solicited and unsolicited adverse event reports.

## 5.10 Stopping rules

If the non-relapse mortality rate in the experimental group receiving high-dose melphalan and bortezomib within the first 28 days after transplantation exceeds 10% then the study will be stopped. Resumption of patient accrual will only be permitted after review of interim results by the Institutional Review Board and the Data Safety Monitoring Board.

# 5.11 Monitoring Compliance.

Patients enrolled into the study will monitored for treatment actually received. Failure to comply with study conditioning regimen would first trigger an intervention to improve compliance.

## 5.12 Data Management and Analysis

Case report forms will be created for management of data collected during this study. A database in Access will be created based on the case report forms. All study data will be imported into SAS and data management will be utilized to flag, and generate queries on out of range data issues until they are resolved. All analysis will be performed using SAS software version 9.2 (SAS Institute Inc. Cary, NC).

## **6.0 Administrative requirements**

#### 6.1 Good Clinical Practice

The study will be conducted in accordance with the International Conference on Harmonisation (ICH) for Good Clinical Practice (GCP) and the appropriate regulatory requirement(s). The investigator will be thoroughly familiar with the appropriate use of the drug as described in the protocol and Investigator's Brochure. Essential clinical documents will be maintained to demonstrate the validity of the study and the integrity of the data collected. Master files should be established at the beginning of the study, maintained for the duration of the study and retained according to the appropriate regulations.

#### 6.2 Ethical Considerations

The study will be conducted in accordance with ethical principles founded in the Declaration of Helsinki. The IRB/IEC will review all appropriate study documentation in order to safeguard the rights, safety and well-being of the patients. The study will only be conducted at sites where IRB/IEC approval has been obtained. The protocol, informed consent, advertisements (if applicable), written information given to the patients (including diary cards), safety updates, annual progress reports, and any revisions to these documents will be provided to the IRB/IEC by the investigator.

## 6.3 Patient Information and Informed Consent

After the study has been fully explained, written informed consent will be obtained from either the patient or his/her guardian or legal representative prior to study participation. The method of obtaining and documenting the informed consent and the contents of the consent will comply with ICH-GCP and all applicable regulatory requirement(s).

A conference will be held with the patient and family to discuss this study and alternative treatments available for treatment of the underlying disease. All potential risks associated with the use of bortezomib, melphalan and HSCT will be discussed as objectively as possible. It will be explained that patients offered this treatment have advanced malignancy with life expectancy of months to no more than 1-2 years with conventional treatments. Informed consent from the patient will be obtained using the IRB-approved consent form describing this protocol. The patient has the right to review and correct the results of the pre-transplant evaluation.

## 6.4 Protocol Registration

All patients will be assigned a unique patient number (UPN) in accordance with HUMC Standard Practice.

## 6.5 Patient Confidentiality

In order to maintain patient privacy, all data capture records, drug accountability records, study reports and communications will identify the patient by initials and the assigned patient number. The patient's confidentiality will be maintained and will not be made publicly available to the extent permitted by the applicable laws and regulations.

#### 6.6 Record Retention

The investigator will maintain all study records according to ICH-GCP and applicable regulatory requirement)s). The licensed medical records department, affiliated with the institution where the patient receives medical card, maintains all original inpatient and outpatient chart documents.

## 6.7 Investigation New Drug Exemption

All of the drugs employed in this protocol are commercially available and an IND exemption is not required for the conduct of this study. The study will be conducted in accordance with current Good Clinical Practice guidelines.

# 7.0 Karnofsky Performance Status Scale

The following table presents the Karnofsy performance status scale<sup>1</sup>:

| Points | Description |
|---|---|
| 100 | Normal, no complaints, no evidence of disease |
| 90 | Able to carry on normal activity |
| 80 | Normal activity with effort; some signs or symptoms of disease |
| 70 | Cares for self; unable to carry on normal activity or to do active work |
| 60 | Requires occasional assistance but is able to care for most of his/her needs |
| 50 | Requires considerable assistance and frequent medical care |
| 40 | Disabled; requires special care and assistance |
| 30 | Severely disabled; hospitalization indicated. Death not imminent |
| 20 | Very sick; hospitalization necessary; active support treatment necessary |
| 10 | Moribund; fatal processes progressing rapidly |
| 0 | Dead |

Mor V, Laliberte L, Morris JN, Wiemann M. The Karnofsky Performance Status Scale: an examination of its reliability and validity in a research setting. *Cancer* 1984;53:2002-2007.

# 8.0 Body Surface Area and Creatinine Clearance Calculations

Body surface area (BSA) should be calculated using a standard nomogram that yields the following results in meters squared (m<sup>2</sup>):

$$BSA = \sqrt{\frac{Ht(inches) \times Wt(lbs)}{3131}}$$

or

$$_{\mathrm{BSA}}=\sqrt{\frac{Ht(cm)\times Wt(kg)}{3600}}$$

Creatinine clearance (CrCl) can be calculated using the Cockroft-Gault equation as follows:

$$CrCl (ml/min) = (140-age) (actual wt in kg)$$
 $72 ext{ x serum creatinine (mg/dl)}$ 

For females use 85% of calculated CrCl value.

Note: In markedly obese patients, the Cockroft-Gault formula will tend to overestimate the creatinine clearance. (Adipose tissue tends to contribute little creatinine requiring renal clearance.) 12.0 New York Heart Association Classification of Cardiac Disease

The following table presents the NYHA classification of cardiac disease:

| Class | Functional Capacity | <b>Objective Assessment</b> |
|---|---|---|
| I | Patients with cardiac disease but without resulting limitations of | No objective evidence |
| | physical activity. Ordinary physical activity does not cause undue | of cardiovascular |
| | fatigue, palpitation, dyspnea, or anginal pain. | disease. |
| II | Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity | Objective evidence of minimal |
| | results in fatigue, palpitation, dyspnea, or anginal pain. | cardiovascular disease. |

| III | Patients with cardiac disease resulting in marked limitation of | Objective evidence of |
|---|---|---|
| | physical activity. They are comfortable at rest. Less than ordinary | moderately severe |
| | activity causes fatigue, palpitation, dyspnea, or anginal pain. | cardiovascular disease. |
| IV | Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased. | Objective evidence of severe cardiovascular disease. |

Source: The Criteria Committee of New York Heart Association. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. 9th Ed. Boston, MA: Little, Brown & Co; 1994:253-256.

#### 9.0 Declaration of Helsinki

#### **World Medical Association Declaration of Helsinki:**

Ethical Principles for Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly Helsinki, Finland, June 1964 and amended by the 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 and the 52nd WMA General Assembly, Edinburgh, Scotland, October 2000

#### INTRODUCTION

- 1. The World Medical Association has developed the Declaration of Helsinki as a statement of ethical principles to provide guidance to physicians and other participants in medical research involving human subjects. Medical research involving human subjects includes research on identifiable human material or identifiable data.
- 2. It is the duty of the physician to promote and safeguard the health of the people. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.
- 3. The Declaration of Geneva of the World Medical Association binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act only in the patient's interest when providing medical care which might have the effect of weakening the physical and mental condition of the patient."
- 4. Medical progress is based on research which ultimately must rest in part on experimentation involving human subjects.
- 5. In medical research on human subjects, considerations related to the well-being of the human subject should take precedence over the interests of science and society.
- 6. The primary purpose of medical research involving human subjects is to improve prophylactic, diagnostic and therapeutic procedures and the understanding of the aetiology and pathogenesis of disease. Even the best proven prophylactic, diagnostic, and therapeutic

- methods must continuously be challenged through research for their effectiveness, efficiency, accessibility and quality.
- 7. In current medical practice and in medical research, most prophylactic, diagnostic and therapeutic procedures involve risks and burdens.
- 8. Medical research is subject to ethical standards that promote respect for all human beings and protect their health and rights. Some research populations are vulnerable and need special protection. The particular needs of the economically and medically disadvantaged must be recognized. Special attention is also required for those who cannot give or refuse consent for themselves, for those who may be subject to giving consent under duress, for those who will not benefit personally from the research and for those for whom the research is combined with care.
- 9. Research Investigators should be aware of the ethical, legal and regulatory requirements for research on human subjects in their own countries as well as applicable international requirements. No national ethical, legal or regulatory requirement should be allowed to reduce or eliminate any of the protections for human subjects set forth in this Declaration.

#### BASIC PRINCIPLES FOR ALL MEDICAL RESEARCH

- 1. It is the duty of the physician in medical research to protect the life, health, privacy, and dignity of the human subject.
- 2. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and on adequate laboratory and, where appropriate, animal experimentation.
- 3. Appropriate caution must be exercised in the conduct of research which may affect the environment, and the welfare of animals used for research must be respected.
- 4. The design and performance of each experimental procedure involving human subjects should be clearly formulated in an experimental protocol. This protocol should be submitted for consideration, comment, guidance, and where appropriate, approval to a specially appointed ethical review committee, which must be independent of the investigator, the sponsor or any other kind of undue influence. This independent committee should be in conformity with the laws and regulations of the country in which the research experiment is performed. The committee has the right to monitor ongoing trials. The researcher has the obligation to provide monitoring information to the committee, especially any serious adverse events. The researcher should also submit to the committee, for review, information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest and incentives for subjects.
- 5. The research protocol should always contain a statement of the ethical considerations involved and should indicate that there is compliance with the principles enunciated in this Declaration.
- 6. Medical research involving human subjects should be conducted only by scientifically qualified persons and under the supervision of a clinically competent medical person. The responsibility for the human subject must always rest with a medically qualified person and never rest on the subject of the research, even though the subject has given consent.

- 7. Every medical research project involving human subjects should be preceded by careful assessment of predictable risks and burdens in comparison with foreseeable benefits to the subject or to others. This does not preclude the participation of healthy volunteers in medical research. The design of all studies should be publicly available.
- 8. Physicians should abstain from engaging in research projects involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians should cease any investigation if the risks are found to outweigh the potential benefits or if there is conclusive proof of positive and beneficial results.
- 9. Medical research involving human subjects should only be conducted if the importance of the objective outweighs the inherent risks and burdens to the subject. This is especially important when the human subjects are healthy volunteers.
- 10. Medical research is only justified if there is a reasonable likelihood that the populations in which the research is carried out stand to benefit from the results of the research.
- 11. The subjects must be volunteers and informed participants in the research project.
- 12. The right of research subjects to safeguard their integrity must always be respected. Every precaution should be taken to respect the privacy of the subject, the confidentiality of the patient's information and to minimize the impact of the study on the subject's physical and mental integrity and on the personality of the subject.
- 13. In any research on human beings, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail. The subject should be informed of the right to abstain from participation in the study or to withdraw consent to participate at any time without reprisal. After ensuring that the subject has understood the information, the physician should then obtain the subject's freely-given informed consent, preferably in writing. If the consent cannot be obtained in writing, the non-written consent must be formally documented and witnessed.
- 14. When obtaining informed consent for the research project the physician should be particularly cautious if the subject is in a dependent relationship with the physician or may consent under duress. In that case the informed consent should be obtained by a well-informed physician who is not engaged in the investigation and who is completely independent of this relationship.
- 15. For a research subject who is legally incompetent, physically or mentally incapable of giving consent or is a legally incompetent minor, the investigator must obtain informed consent from the legally authorized representative in accordance with applicable law. These groups should not be included in research unless the research is necessary to promote the health of the population represented and this research cannot instead be performed on legally competent persons.
- 16. When a subject deemed legally incompetent, such as a minor child, is able to give assent to decisions about participation in research, the investigator must obtain that assent in addition to the consent of the legally authorized representative.
- 17. Research on individuals from whom it is not possible to obtain consent, including proxy or

advance consent, should be done only if the physical/mental condition that prevents obtaining informed consent is a necessary characteristic of the research population. The specific reasons for involving research subjects with a condition that renders them unable to give informed consent should be stated in the experimental protocol for consideration and approval of the review committee. The protocol should state that consent to remain in the research should be obtained as soon as possible from the individual or a legally authorized surrogate.

18. Both authors and publishers have ethical obligations. In publication of the results of research, the investigators are obliged to preserve the accuracy of the results. Negative as well as positive results should be published or otherwise publicly available. Sources of funding, institutional affiliations and any possible conflicts of interest should be declared in the publication. Reports of experimentation not in accordance with the principles laid down in this Declaration should not be accepted for publication.

# ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 1. The physician may combine medical research with medical care, only to the extent that the research is justified by its potential prophylactic, diagnostic or therapeutic value. When medical research is combined with medical care, additional standards apply to protect the patients who are research subjects.
- 2. The benefits, risks, burdens and effectiveness of a new method should be tested against those of the best current prophylactic, diagnostic, and therapeutic methods. This does not exclude the use of placebo, or no treatment, in studies where no proven prophylactic, diagnostic or therapeutic method exists.
- 3. At the conclusion of the study, every patient entered into the study should be assured of access to the best proven prophylactic, diagnostic and therapeutic methods identified by the study.
- 4. The physician should fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study must never interfere with the patient-physician relationship.
- 5. In the treatment of a patient, where proven prophylactic, diagnostic and therapeutic methods do not exist or have been ineffective, the physician, with informed consent from the patient, must be free to use unproven or new prophylactic, diagnostic and therapeutic measures, if in the physician's judgment it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, these measures should be made the object of research, designed to evaluate their safety and efficacy. In all cases, new information should be recorded and, where appropriate, published. The other relevant guidelines of this Declaration should be followed.

# 10.0Common Terminology Criteria for Adverse Events 3.0

http://ctep.cancer.gov/reporting/ctc.html

#### 11.0 References

Adams J, Palombella VJ, Sausville EA, Johnson J, Destree A, Lazarus DD et al. Proteasome inhibitors: a novel class of potent and effective antitumor agents. Cancer Res 1999; 59 (11):2615-22.

Aghajanian C, Dizon DS, Sabbatini P, et al. Phase I trial of bortezomib and carboplatin in recurrent ovarian or primary peritoneal cancer. J Clin Oncol 2005;23:5943-49

Alexanian R, Dimopoulos M. The treatment of multiple myeloma. N Engl J Med. 1994;330:484-489

Attal M, Huguet F, Schlaifer D, et al. Intensive combination therapy for previously untreated aggressive myeloma. Blood 1992;79:1130-6

Attal M, Harousseau J-L, Stoppa A-M, et al. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. N Engl J Med 1996;335:91-7

Attal M, Harousseau JL, Facon T, et al. Single versus double autologous stem-cell transplantation for multiple myeloma. N Engl J Med. 2003;349:2495-502

Badros A. Barlogie B, Siegel E. et al. Results of autologous stem cell transplant in multiple myeloma patients with renal failure. Br J Haematol 2001;114:822-9

Barlogie B, Jagannath S, Vesole DH, et al. Superiority of tandem autologous transplantation over standard therapy for previously untreated multiple myeloma. Blood 1997;89:789-93

Barlogie B, Kyle RA, Anderson KC, et al. Standard chemotherapy compared with high-dose chemoradiotherapy for multiple myeloma: final results of phase III US Intergroup Trial S9321. J Clin Oncol 2006;24:929-36

Berenson JR, Yang HH, Sadler K, et al. Phase I/II trial assessing bortezomib and melphalan combination therapy for the treatment of patients with relapsed or refractory multiple myeloma. J Clin Oncol 2006;24:937-44

Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G et al. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol 1998; 102 (5):1115-23.

Blade J, Rosinol L, Sureda A, et al. High-dose therapy intensification compared with continued standard chemotherapy in multiple myeloma patients responding to the initial chemotherapy: long-term results from a prospective randomized trial from the Spanish cooperative group PETHEMA. Blood 2005;106:3755-9

Child JA, Morgan GJ, Davies FE, et al. High-dose chemotherapy with hematopoietic stem-cell rescue for multiple myeloma. N Engl J Med. 2003; 348:1875-83

Cleveland, WS: Robust locally-weighted regression and smoothing scatterplots. J. Am Stat Assoc. 1979; 74: 829-836

Cox, DR. Regression models and life tables (with discussion). J R Stat Soc B.1972; 34:187-220. Cusack JC, Jr., Liu R, Houston M, Abendroth K, Elliott PJ, Adams J et al. Enhanced chemosensitivity to CPT-11 with proteasome inhibitor PS-341: implications for systemic nuclear factor-kappaB inhibition. Cancer Res 2001; 61 (9):3535-40.

Desikan R, Barlogie B, Sawyer J, et al. Results of high dose therapy for 1000 patients with multiple myeloma: durable complete remission and superior survival in the absence of chromosome 13 abnormalities. Blood 2000;95:4008-10

Dixon, DO. and Simon, R. Sample size considerations for studies comparing survival curves using historical controls, J Clin Epidemiol. 1988; 41: 1209-1213.

Durie BG. Kyle RA. Belch A, et al. Myeloma management guidelines: a consensus report from the Scientific Advisors of the International Myeloma Foundation. Hematol J 2003;4:379-98

Fassas AB, Barlogie B, Ward S, et al. Survival after relapse following tandem autotransplants in multiple myeloma patients: The University of Arkansas total therapy I experience. Br J Haematol 2003;123:484-9

Fermand JP, Ravaud P, Chevret S, et al. High-dose therapy and autologous peripheral blood stem cell transplantation in multiple myeloma: up-front or rescue treatment? Results of a multicenter sequential randomized clinical trial. Blood 1998;92:3131-6

Fermand JP, Katsahian S, Devine M, et al. High-dose therapy and autologous blood stem-cell transplantation compared with conventional treatment in myeloma patients aged 55 to 65 years: long-term results of a randomized control trial from the Group Myelome-Autogreffe. J Clin Oncol 2005;23:9227-33

Fonseca R, Barlogie B, Bataille R, et al. Genetics and cytogenetics of multiple myeloma; a workshop report. Cancer Res 2004;64:1546-58

Fossella FV, DeVore R, Kerr RN, Crawford J, Natale RR, Dunphy F et al. Randomized phase III trial of docetaxel versus vinorelbine or ifosfamide in patients with advanced non-small-cell lung cancer previously treated with platinum-containing chemotherapy regimens. The TAX 320 Non-Small Cell Lung Cancer Study Group. J Clin Oncol 2000; 18 (12):2354-62.

Fossella F. Docetaxel + Cisplatin (DC) and Docetaxel + Carboplatin (DCb) vs Vinorelbine + Cisplatin (VC) in chemotherapy-naïve patients with advanced and metastatic non-small cell lung cancer (NSCLC): Results of a multicenter, randomized phase III study. European Journal of Cancer, European Cancer Conference, ECCO 11, 2001; Lisbon, Portugal. 37(suppl 6):S154. Abstract 562

Gharton G, Svensson H, Bjorkstrand B, et al. Syngeneic transplantation in multiple myeloma – a case-matched comparison with autologous and allogeneic transplantation. European Group for Blood and Marrow Transplantation. Bone Marrow Transpl 1999;24:741-5

Goldberg SL, Klumpp TR, Magdalinski AJ, Mangan KF. Value of the pretransplant evaluation in predicting toxic day-100 mortality among blood stem-cell and bone marrow transplant recipients. J Clin Oncol 1998;16:3796-802

Gouyette A, Hartmann O, Pico J-L. Pharmacokinetics of high-dose melphalan in children and adults. Cancer Chemother Pharmacol 1986;16:184-9

Hall AG, Tilby MJ. Mechanisms of action of, and modes of resistance to, alkylating agents used in the treatment of hematological malignancies. Blood Rev 1992;6:163-73

Harousseau JL, Attal M, Divine M, et al. Autologous stem cell transplantation after first remission induction treatment in multiple myeloma: a report of the French Registry on autologous transplantation in multiple myeloma. Blood 1995;85:3077-85

Hideshima T, Richardson P, Chauhan D, Palombella VJ, Elliott PJ, Adams J et al. The proteasome inhibitor PS-341 inhibits growth, induces apoptosis, and overcomes drug resistance in human multiple myeloma cells. Cancer Res 2001; 61 (7):3071-6.

Hollmig K, Stover J, Talamo G, et al. Addition of bortezomib (Velcade<sup>TM</sup>) to high dose melphalan (VelMel) as an effective conditioning regimen with autologous stem cell support in multiple myeloma (MM). Blood 2004;104:266a

Jagannath S, Barlogie B, Berenson J et al. A Phase 2 study of two doses of bortezomib in relapsed or refractory myeloma. Br J Haematol 2004: 127:165-172

Kergueris MF, Milpied N, Moreau P, et al. Pharmacokinetics of high-dose melphalan in adults: Influence of renal function. Anticancer Res 1994;14:2379-82

LeBlanc R, Catley LP, Hideshima T, Lentzsch S, Mitsiades CS, Mitsiades N et al. Proteasome inhibitor PS-341 inhibits human myeloma cell growth in vivo and prolongs survival in a murine model. Cancer Res 2002; 62 (17):4996-5000.

Lee CK, Barlogie B, Zangari M, et al. Transplantation as salvage therapy for high-risk patients with myeloma in relapse. Bone Marrow Transpl 2002;30:873-8

Lightcap ES, McCormack TA, Pien CS, Chau V, Adams J, Elliott PJ. Proteasome inhibition measurements: clinical application. Clin Chem 2000; 46 (5):673-83.

McConkey DJ, Pettaway C, Elliott P, Adam J, Papandreou C, Herrmann JL et al. The proteasome as a new drug target in metastatic prostate cancer. 7th Annual Genitourinary Oncology Conference, 1999; Houston, TX. Abstract

McElwain TJ, Powles RL. High-dose intravenous melphalan for plasma-cell leukaemia and myeloma. Lancet 1983;2(8354):822-4

Mehta J, Tricot G, Jagannath S, et al. Salvage autologous or allogeneic transplantation for multiple myeloma refractory to or relapseing after a first-line autograft? Bone Marrow Transpl 1998;21:887-92

Mitsiades N, Mitsiades CS, Richardson PG, et al. The proteasome inhibitor PS-341 potentiates sensitivity of multiple myeloma cells to conventional chemotherapeutic agents: therapeutic applications. Blood 2003;101:2377-80

Nathans D, Fahey JL, Potter M. The formation of myeloma protein by a mouse plasma cell tumor. J Exp Med 1958;108:121-30

Orlowski RZ, Stinchcombe TE, Mitchell BS, Shea TC, Baldwin AS, Stahl S et al. Phase I Trial of the Proteasome Inhibitor PS-341 in Patients with Refractory Hematologic Malignancies. J Clin Oncol 2002; 20 (22):4420-7.

Orlowski RZ, Voorhees PM, Garcia RA, et al. Phase I trial of the proteasome inhibitor bortezomib and pegylated liposomal doxorubicin in patients with advanced hematologic malignancies. Blood 2005;105:3058-65

Paccagnella A, Chiarion-Sileni V, Soesan M, et al. Second and third responses to the same induction regimen in relapsing patients with multiple myeloma. Cancer 1991;68:975-80

Palumbo A, Bringhen S, Petrucci MT, et al. Intermediate-dose melphalan improves survival of myeloma patients aged 50 to 70: results of a randomized controlled trial. Blood 2004;104:3052-7

Pandit S, Vesole DH. Relapsed multiple myeloma. Curr Treat Options Oncol 2001;2:261-9 Papandreou C, Daliani D, Millikan RE, Tu S, Pagliaro L, Adam J. Phase I Study of Intravenous (I.V.) Proteasome Inhibitor PS-341 in Patients (Pts) with Advanced Malignancies. Proc Am Soc Clin Oncol, 2001. Abstract 340

Pineda-Roman M, Fox MH, Hollmig KA, et al. Retrospective analysis of fractionated high-dose melphalan (F-Mel) and bortezomib-thalidomide-dexamethasone (VTD) with autotransplant (AT) support for advanced and refractory multiple myeloma (AR-MM). Blood 2006;108:884a

Pinguet F, Martel P, Fabbro M, et al. Pharmacokinetics of high-dose intravenous melphalan in patients undergoing peripheral blood hematopoietic progenitor-cell transplantation. Antican Res 1997;17:605-12

Pink MM, Pien CS, Ona VO, Worland P, Adams J, Kauffman MG. PS-341 enhances chemotherapeutic effect in human xenograft models. Proc Am Assoc Cancer Res, 2002; San Francisco, CA. Abstract 787

Reece PA, Hill HS, Green RM, et al. Renal clearance and protein binding of melphalan in patients with cancer. Cancer Chemother Pharmacol 1988;22:348-52

Richardson PG, Barlogie B, Berenson J et al. A Phase II study of Bortezomib in Relapsed, Refractory Myeloma. N Engl J Med 2003; 348:2609-2617

Richardson PG, et al., Bortezomib or High-Dose Dexamethasone for Relapsed Multiple Myeloma. N Engl J Med 2005; 352:2487-98.

Richardson et al, Bortezomib Continues to Demonstrate Superior Efficacy Compared With High-Dose Dexamethasone in Relapsed Multiple Myeloma: Updated Results of the APEX Trial. Blood, 2005; 106: Abstract 2547.

Richardson et al. Multicenter, phase I, dose-escalation trial of lenalidomide plus bortezomib for relapsed zand relapsed/refractory multiple myeloma. J Clion Oncol. 2009 Sep 28. [Epub ahead of print].

Rowley SD, Siegel, D, Donato ML, et al. Combination melphalan and bortezomib conditioning with autologous hematopoeitic stem cell support in patients with advanced multiple myeloma. A phase I/II study. Blood 2009;114:499

Samuels BL, Bitran JD. High-dose intravenous melphalan: A review. J Clin Oncol 1995;13:1786-99

Siegel DS, Desikan KR, Mehta J, et al. Age is not a prognostic variable with autotransplants for multiple myeloma. Blood 1999;93:51-54

Spanswick VJ, Craddock C, Sekhar M, et al. Repair of DNA interstrand crosslinks as a mechanism of clinical resistance to melphalan in multiple myeloma. Blood 2002;100:224-9

Steiner P, Neumeier H, Lightcap E, Sadis S, Pien C, Pink M et al. Adaptation of Human Tumor Cell Lines to PS-341. AACR-NCI-EORTC International Conference, 2001; Miami Beach, FL. Millennium Pharmaceuticals, Inc., 75 Sidney Street, Cambridge, MA 02139. Abstract

Teicher BA, Ara G, Herbst R, Palombella VJ, Adams J. The proteasome inhibitor PS-341 in cancer therapy. Clin Cancer Res 1999; 5 (9):2638-45.

Therneau, TM. and Grambsch, P. Modeling Survival Data. New York, NY: Springer, 2000.

Tricot G, Jagannath S, Vesoled DH, Crowley J, Barlogie B. Relapse of multiple myeloma after autologous transplantation: survival after salvage therapy. Bone Marrow Transpl 1995;16:7-11

Tricot G, Alberts DS, Johnson C, et al. Safety of autotransplants with high-dose melphalan in renal failure: a pharmacokinetic and toxicity study. Clin Ca Res 1996;2:947-52

Tricot G, Spencer T, Sawyer J, et al. Predicting long-term (≥5 years) event-free survival in multiple myeloma patients following planned tandem autotransplants. Br J Haematol 2002;116:211-7

VELCADE (bortezomib) [package insert]. Cambridge, MA: Millennium Pharmaceuticals, Inc.; 2003.

Vesole D, Barlogie B, Jagannath S, et al. High dose chemotherapy for refractory multiple myeloma: improved prognosis with better supportive care and double transplants. Blood 1994:84:950-6